CLINICAL TRIAL: NCT02278341
Title: A Phase 3, Randomized, Open-Label, Active-Controlled Study to Evaluate the Efficacy and Safety of Roxadustat in the Maintenance Treatment of Anemia in End Stage Renal Disease Patients on Stable Dialysis
Brief Title: Roxadustat in the Treatment of Anemia in End Stage Renal Disease (ESRD) Patients on Stable Dialysis
Acronym: Pyrenees
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Astellas Pharma Europe B.V. (Industry)
Collaborators: Kyntra Bio (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1517-CL-0613; 2013-001497-16 (EudraCT Number)
Record Dates: First submitted 2014-10-28; First posted 2014-10-30 (Estimated); Results first posted 2020-08-26 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-11

CONDITIONS: Anemia; End Stage Renal Disease (ESRD)
Keywords: ASP1517; FG-4592; Anemia; End Stage Renal Disease (ESRD); Erythropoetin Stimulating Agents (ESAs); Chronic Kidney Disease; Hematopoetic Agents; HIF-PH inhibitor; Hemoglobin; Dialysis; roxadustat
MeSH Terms: conditions — Anemia; Kidney Failure, Chronic; Renal Insufficiency, Chronic | interventions — roxadustat; Epoetin Alfa; Darbepoetin alfa; Iron

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Roxadustat (Experimental): Participants received roxadustat three times a week (TIW) for at least 52 weeks up to a maximum of 104 weeks. Participants received initial dose of roxadustat in doses of 100 mg, 150 mg or 200 mg, according to the average weekly dose of epoetin or darbepoetin alfa prior to randomization. Participants' roxadustat dosage was adjusted every 4 weeks to maintain Hb level within the target range 10.0 to 12.0 g/dL. Dose adjustment steps were as follows: 20, 40, 50, 70, 100, 150, 200, 250, 300, and 400 mg. Oral iron treatment of 200 mg was allowed for supplementation to support erythropoiesis. Treatment with intravenous iron was allowed only if certain protocol criteria were met.
  Interventions: Drug: Roxadustat; Drug: Iron
- ESA (Erythropoiesis Stimulating Agent) treatment (Active Comparator): Participants received epoetin alfa once weekly, twice weekly or TIW and darbepoetin alfa once a week or once every other week. Participants were treated for at least 52 weeks up to a maximum of 104 weeks. Treatment dosage was adjusted according to the pre-specified rule of keeping the participant's Hb levels between 10.0 to 12.0 g/dL. Participants were not allowed to switch from the epoetin alfa to darbepoetin alfa or vice versa.
  Interventions: Drug: Epoetin alfa; Drug: Darbepoetin alfa; Drug: Iron

INTERVENTIONS:
Drug: Roxadustat — Participants received initial dose of roxadustat orally as a tablet in doses of 100 mg, 150 mg or 200 mg, according to the average weekly dose of epoetin or darbepoetin alfa prior to randomization. Participants' roxadustat dosage was adjusted every 4 weeks to maintain Hb level within the target range 10.0 to 12.0 g/dL. Dose adjustment steps were as follows: 20, 40, 50, 70, 100, 150, 200, 250, 300, and 400 mg. Oral iron treatment of 200 mg was allowed for supplementation to support erythropoiesis. Treatment with intravenous iron was allowed only if certain protocol criteria were met.
  Other Names: ASP1517; FG-4592
  Arms: Roxadustat
Drug: Epoetin alfa — Participants received epoetin alfa via intravenous or subcutaneous injection, once a week, twice a week, or three times a week (TIW). Epoetin alfa dosage was adjusted to maintain Hb level within the target range. Dosing of epoetin alfa was per UK SmPC of Eprex®. Participants received IV iron supplementation according to the standard of care.
  Other Names: Eprex
  Arms: ESA (Erythropoiesis Stimulating Agent) treatment
Drug: Darbepoetin alfa — Participants received darbepoetin alfa via intravenous or subcutaneous injection, once a week or once every other week. Darbepoetin alfa dosage was adjusted to maintain Hb level within the target range. Dosing of darbepoetin alfa was per EU SmPC of Aranesp®. Participants received IV iron supplementation according to the standard of care.
  Other Names: Aranesp
  Arms: ESA (Erythropoiesis Stimulating Agent) treatment
Drug: Iron — Oral iron treatment was recommended for supplementation to support erythropoiesis and as first-line treatment for iron deficiency, unless participant was intolerant to this treatment. For participants receiving roxadustat the recommended daily dose was 200 mg of elemental iron. Participants were advised to take roxadustat at least 1 hour before or 1 hour after oral iron. Intravenous iron supplementation for participants receiving roxadustat was allowed if all of the following criteria were met: The participant's Hb level had not responded adequately to roxadustat following two consecutive dose increases or reached the maximum dose limit, and participant's ferritin was < 100 ng/mL (< 220 pmol/L) or TSAT < 20%, or the participant was intolerant of oral iron therapy. For participants treated with epoetin alfa or darbepoetin alfa, IV iron supplementation was given according to standard of care.

SUMMARY:
This study was conducted to explore a new therapy for anemia in participants with end stage renal disease (ESRD) on dialysis. Anemia is a reduced number of red blood cells or hemoglobin. Hemoglobin (which contains iron) is important for the transport of oxygen in your blood. The purpose of this study was to evaluate if roxadustat is effective and safe in the maintenance treatment of anemia in ESRD participants on stable dialysis. Roxadustat was compared to epoetin alfa and darbepoetin alfa, commercially available medicines for treatment of anemia.

DETAILED DESCRIPTION:
This study consisted of three study periods as follows:

* Screening Period: up to 6 weeks
* Treatment Period: a minimum of 52 weeks up to a maximum of 104 weeks
* Follow-up Period: 4 weeks

ELIGIBILITY:
Inclusion Criteria:

Main Inclusion:

* Participant is on stable hemodialysis (HD), hemodiafiltration (HDF) or peritoneal dialysis (PD) treatment with the same mode of dialysis for ≥4 months prior to randomization.
* Participant is on IV or SC epoetin or IV or SC darbepoetin alfa treatment for ≥8 weeks prior to randomization with stable weekly doses (during 4 weeks prior to randomization).
* Mean of the participant's three most recent Hb values, as measured by central laboratory, during the Screening Period.
* Participant's alanine aminotransferase (ALT) and aspartate aminotransferase (AST) are ≤3 x upper limit of normal (ULN), and total bilirubin (TBL) is ≤1.5 x ULN

Exclusion Criteria:

Main Exclusion:

* Participant has received a red blood cell (RBC) transfusion within 8 weeks prior to randomization.
* Participant has a known hereditary hematologic disease such as thalassemia or sickle cell anemia, pure red cell aplasia, or other known causes for anemia other than Chronic Kidney Disease (CKD).
* Participant has had a myocardial infarction, acute coronary syndrome, stroke, seizure, or a thrombotic/thrombo-embolic event (e.g., deep vein thrombosis or pulmonary embolism) within 12 weeks prior to randomization.
* Participant has had uncontrolled hypertension, in the opinion of the investigator, within 2 weeks prior to randomization.
* Participant has a history of malignancy, except for the following: cancers determined to be cured or in remission for ≥5 years, curatively resected basal cell or squamous cell skin cancers, cervical cancer in situ, or resected colonic polyps.
* Participant has had any prior organ transplant (that has not been explanted), or participant is scheduled for organ transplantation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 838 (Actual)
Dates: Start 2014-11-21 (Actual); Primary Completion 2017-06-08 (Actual); Study Completion 2018-07-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Physician, Study Director — Astellas Pharma Europe B.V.
Locations (143):
- Belgium (9):
  - Site BE32004, Brussels, Flemish Brabant
  - Site BE32001, Aalst
  - Site BE32019, Antwerp
  - Site BE32002, Antwerp
  - Site BE32012, Baudour
  - Site BE32017, Bonheiden
  - Site BE32003, Leuven
  - Site BE32013, Liège
  - Site BE32011, Roeselare
- Bulgaria (15):
  - Site BG35925, Blagoevgrad
  - Site BG35931, Haskovo
  - Site BG35915, Pleven
  - Site BG35909, Plovdiv
  - Site BG35919, Plovdiv
  - Site BG35920, Rousse
  - Site BG35938, Shumen
  - Site BG35924, Sofia
  - Site BG35906, Sofia
  - Site BG35921, Sofia
  - Site BG35907, Stara Zagora
  - Site BG35916, Varna
  - Site BG35918, Varna
  - Site BG35903, Veliko Tarnovo
  - Site BG35937, Yambol
- Croatia (7):
  - Site HR38509, Zagreb, City of Zagreb
  - Site HR38508, Čakovec
  - Site HR38505, Karlovac
  - Site HR38507, Osijek
  - Site HR38506, Rijeka
  - Site HR38504, Slavonski Brod
  - Site HR38501, Zadar
- Czechia (3):
  - Site CZ42008, Liberec
  - Site CZ42021, Prague
  - Site CZ42015, Rakovník
- France (5):
  - Site FR33005, Amiens
  - Site FR33010, La Tronche
  - Site FR33007, Saint Priez En Jarez
  - Site FR33055, Saint-Ouen
  - Site FR33056, Valenciennes
- Georgia (3):
  - Site GE99503, Tbilisi
  - Site GE99504, Tbilisi
  - Site GE99508, Tbilisi
- Germany (12):
  - Site DE49056, Dormagen, North Rhine-Westphalia
  - Site DE49067, Berlin
  - Site DE49073, Cloppenburg
  - Site DE49008, Dresden
  - Site DE49054, Düsseldorf
  - Site DE49020, Frankfurt am Main
  - Site DE49065, Hamburg
  - Site DE49075, Heilbronn
  - Site DE49001, Kaiserslautern
  - Site DE49070, München
  - Site DE49002, Solingen
  - Site DE49071, Villingen-Schwenningen
- Hungary (12):
  - Site HU36033, Baja
  - Site HU36036, Esztergom
  - Site HU36031, Győr
  - Site HU36026, Kaposvár
  - Site HU36027, Kistarcsa
  - Site HU36032, Pécs
  - Site HU36035, Pécs
  - Site HU36034, Salgótarján
  - Site HU36004, Szeged
  - Site HU36046, Székesfehérvár
  - Site HU36006, Szombathely
  - Site HU36003, Zalsaegerszeg
- Italy (12):
  - Site IT39028, Prato, Frazione Di Galciana
  - Site IT39039, Cremona, Lombardy
  - Site IT39014, Mestre, Venezia
  - Site IT39010, Brescia
  - Site IT39008, Lecco
  - Site IT39006, Milan
  - Site IT39037, Modena
  - Site IT39022, Padua
  - Site IT39036, Pavia
  - Site IT39005, Roma
  - Site IT39035, Torino
  - Site IT39032, Trieste
- Poland (7):
  - Site PL48002, Katowice
  - Site PL48001, Krakow
  - Site PL48013, Szczecin
  - Site PL48005, Warsaw
  - Site PL48006, Wroclaw
  - Site PL48009, Wroclaw
  - Site PL48014, Zamość
- Portugal (8):
  - Site PT35121, Almada
  - Site PT35127, Aveiro
  - Site PT35139, Cascais
  - Site PT35117, Faro
  - Site PT35128, Gaeiras
  - Site PT35114, Leiria
  - Site PT35102, Porto
  - Site PT35122, Setúbal
- Romania (5):
  - Site RO40018, Bucharest
  - Site RO40003, Bucharest
  - Site RO40015, Bucharest
  - Site RO40019, Bucharest
  - Site RO40004, Oradea
- Russia (14):
  - Site RU70008, Kaluga
  - Site RU70051, Moscow
  - Site RU70005, Moscow
  - Site RU70003, Nizhny Novgorod
  - Site RU70004, Omsk
  - Site RU70014, Rostov-on-Don
  - Site RU70072, Saint Petersburg
  - Site RU70011, Saint Petersburg
  - Site RU70002, Saint Petersburg
  - Site RU70030, Saint Petersburg
  - Site RU70050, Saint Petersburg
  - Site RU70006, Smolensk
  - Site RU70037, Volgograd
  - Site RU70001, Yaroslavl
- Serbia (7):
  - Site RS38102, Belgrade
  - Site RS38105, Belgrade
  - Site RS38120, Belgrade
  - Site RS38104, Belgrade
  - Site RS38117, Kruševac
  - Site RS38101, Niš
  - Site RS38116, Zrenjanin
- Slovakia (5):
  - Site SK42102, Košice
  - Site SK42119, Levice
  - Site SK42120, Lučenec
  - Site SK42113, Púchov
  - Site SK42116, Senica
- Spain (11):
  - Site ES34041, Santiago de Compostela, A Coruna
  - Site ES34009, El Ejido, Almeria
  - Site ES34010, Alcorcón, Madrid
  - Site ES34030, Majadahonda, Madrid
  - Site ES34011, Galdakao, Vizcaya
  - Site ES34002, Badalona-Barcelona
  - Site ES34008, Barcelona
  - Site ES34006, Barcelona
  - Site ES34017, Jaén
  - Site ES34037, Madrid
  - Site ES34052, Valencia
- United Kingdom (8):
  - Site GB44087, Brighton, EastSussex
  - Site GB44011, Canterbury, Kent
  - Site GB44080, Stoke-on-Trent, Staffordshire
  - Site GB44008, Cambridge
  - Site GB44010, Hull
  - Site GB44081, Leicester
  - Site GB44079, Liverpool
  - Site GB44001, Swansea

IPD SHARING:
Plan to Share IPD: Yes
Access to anonymized individual participant level data collected during the study, in addition to study-related supporting documentation, is planned for studies conducted with approved product indications and formulations, as well as products terminated during development. Studies conducted with product indications or formulations that remain active in development are assessed after study completion to determine if Individual Participant Data can be shared. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Access to participant level data is offered to researchers after publication of the primary manuscript (if applicable) and is available as long as Astellas has legal authority to provide the data.
Access Criteria: Researchers must submit a proposal to conduct a scientifically relevant analysis of the study data. The research proposal is reviewed by an Independent Research Panel. If the proposal is approved, access to the study data is provided in a secure data sharing environment after receipt of a signed Data Sharing Agreement.
URL: https://www.clinicaltrials.astellas.com/transparency/

REFERENCES:
- [Derived] Hamano T, Yamaguchi Y, Goto K, Martin S, Jiletcovici A, Dellanna F, Akizawa T, Barratt J. Risk Factors for Thromboembolic Events in Patients With Dialysis-Dependent CKD: Pooled Analysis of Four Global Roxadustat Phase 3 Trials. Adv Ther. 2024 Apr;41(4):1553-1575. doi: 10.1007/s12325-023-02728-2. Epub 2024 Feb 16. PMID 38363466
- [Derived] Natale P, Palmer SC, Jaure A, Hodson EM, Ruospo M, Cooper TE, Hahn D, Saglimbene VM, Craig JC, Strippoli GF. Hypoxia-inducible factor stabilisers for the anaemia of chronic kidney disease. Cochrane Database Syst Rev. 2022 Aug 25;8(8):CD013751. doi: 10.1002/14651858.CD013751.pub2. PMID 36005278
- See also: Link to results on Astellas Clinical Study Results website — https://astellasclinicalstudyresults.com/study.aspx?ID=364

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study population consisted of participants with end-stage renal disease (ESRD) who were on stable hemodialysis (HD) or peritoneal dialysis (PD), and were also on stable treatment with epoetin (i.e. epoetin alfa, beta, theta, zeta, delta or omega) or darbepoetin alfa for anemia.
Pre-assignment Details: Participants were randomized in a 1:1 ratio to roxadustat or ESA (epoetin alfa or darbepoetin alfa). Randomization was stratified by 5 factors: previous ESA treatment, region, history of cardiovascular, cerebrovascular or thromboembolic diseases, average weekly ESA dose 4 weeks prior to randomization and the screening hemaglobin (Hb) value.
Groups:
- ESA (Erythropoiesis-Stimulating Agent): Participants received epoetin alfa once weekly, twice weekly or TIW and darbepoetin alfa once a week or once every other week. Participants were treated for at least 52 weeks up to a maximum of 104 weeks. Treatment dosage was adjusted according to the pre-specified rule of keeping the participant's Hb levels between 10.0 to 12.0 g/dL. Participants were not allowed to switch from epoetin alfa to darbepoetin alfa or vice versa.
Period: Overall Study
Arm/Group | Roxadustat | ESA (Erythropoiesis-Stimulating Agent)
Started | 415 | 421
Received Treatment | 414 | 420
Completed | 297 | 329
Not Completed | 118 | 92
Not completed — Randomized but never received study drug | 1 | 1
Not completed — Adverse Event | 3 | 0
Not completed — Death | 68 | 56
Not completed — Withdrawal by Subject | 30 | 19
Not completed — Lost to Follow-up | 0 | 1
Not completed — Physician Decision | 1 | 1
Not completed — Miscellaneous | 15 | 14

BASELINE CHARACTERISTICS:
Population: The analysis population was the All Randomized, which consisted of participants who were randomized into the study and had the available data.
Groups:
- Total: Total of all reporting groups
Arm/Group | Roxadustat | ESA (Erythropoiesis-Stimulating Agent) | Total
Number analyzed (Participants) | 415 | 421 | 836
Age, Continuous [Mean (Standard Deviation); unit: Years] — Population: The analysis population was the All Randomized population.
  Years | 61 (13.8) | 61.8 (13.4) | 61.4 (13.6)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: The analysis population was the All Randomized population.
  Participants
    Female | 169 | 185 | 354
    Male | 246 | 236 | 482
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: The analysis population was the All Randomized population.
  Participants
    WHITE | 405 | 408 | 813
    BLACK OR AFRICAN AMERICAN | 6 | 6 | 12
    ASIAN | 2 | 3 | 5
    OTHER | 2 | 4 | 6
Baseline Hemoglobin (Hb) Value [Count of Participants; unit: Participants] — Population: The analysis population was the All Randomized population.
  Participants
    <=11.0 g/dL | 267 | 266 | 533
    >11.0 g/dL | 148 | 155 | 303
Baseline Mean Hb [Mean (Standard Deviation); unit: g/dL] — Baseline Hb was defined as the mean of four latest central laboratory Hb values prior or on the same date as first study drug intake (pre-dose). Population: The analysis population was the All Randomized population.
  g/dL | 10.75 (0.62) | 10.77 (0.62) | 10.76 (0.62)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline (BL) to the Average Hemoglobin (Hb) in Weeks 28-36 Without Rescue Therapy [EU (EMA)]
Description: Baseline Hb was defined as the mean of four central laboratory Hb values; four latest Hb values prior or on the same date as the first study drug intake. For participants who did not have an available Hb value during the week 28-36 period, imputation rules were applied. For analyses without rescue therapy, participants who used rescue therapy after the initiation of rescue therapy were set to missing for 6 weeks from the start date of rescue therapy. If no Hb value was available, an imputation technique was used, with the mean of all available values from Day 1 to minimum (End of Efficacy Emergent Period) carried forward.
Time Frame: Baseline and weeks 28 to 36
Population: The analysis population was the Per Protocol Set (PPS) which consisted of all Full Analysis Set (FAS) participants who did not meet any of exclusion criteria from the PPS. The FAS consisted of all randomized participants who received at least one dose of study drug and had at least one post-dose valid Hb assessment.
Measure: Least Squares Mean (95% Confidence Interval); unit: g/dL
Arm/Group | Roxadustat | ESA (Erythropoiesis-Stimulating Agent)
Number analyzed (Participants) | 354 | 381
g/dL | 0.428 [0.350 to 0.506] | 0.193 [0.117 to 0.268]
Statistical Analysis 1: Comparison: Roxadustat vs ESA (Erythropoiesis-Stimulating Agent); The model includes treatment arm, region, CV History, previous ESA treatment, visits and visit by treatment as categorical variables and baseline Hb and baseline Hb by visit as continuous variable; Test type: Non-Inferiority — Non Inferiority, Margin = -0.75; p < 0.001, Mixed Models Analysis — p-value for non-inferiority test based on 1-sided significance level; LSM Difference = 0.235, 95% CI 2-sided [0.132 to 0.339]

2. Primary Outcome: Change From BL to the Average Hb in Weeks 28 to 52 Regardless of Rescue Therapy [US (FDA)]
Description: Baseline Hb was defined as the mean of four central laboratory Hb values: four latest Hb values prior or on the same date as first study drug intake. Change from baseline to the average Hb are observed values. Missing hemoglobin data was imputed for each treatment relying on non-missing data from all participants within each treatment group using the Monte Carlo Markov Chain (MCMC) imputation model with treatment, baseline hemoglobin, randomization stratification factors and the available non missing hemoglobin for each scheduled week.
Time Frame: Baseline and weeks 28 to 52
Population: The analysis population was the All Randomized, which consisted of participants who received at least one dose of study drug, and who had available data.
Measure: Least Squares Mean (95% Confidence Interval); unit: g/dL
Arm/Group | Roxadustat | ESA (Erythropoiesis-Stimulating Agent)
Number analyzed (Participants) | 413 | 420
g/dL | 0.363 [0.288 to 0.438] | 0.192 [0.121 to 0.262]
Statistical Analysis 1: Comparison: Roxadustat vs ESA (Erythropoiesis-Stimulating Agent); The model includes treatment arm, region, CV History, previous ESA treatment as categorical variables and baseline Hb as continuous variable. Statistical analysis used was ANCOVA model with multiple imputations (MI). Missing hemoglobin data was imputed for each treatment relying on non-missing data from all participants within each treatment group using the MCMC imputation model; Test type: Non-Inferiority — Non-Inferiority, Margin = -0.75; p < 0.001, ANCOVA — p-value for non-inferiority test based on 1-sided significance level; LSM Difference = 0.171, 95% CI 2-sided [0.082 to 0.261]

3. Secondary Outcome: Percentage of Participants With Hb Response During Weeks 28 to 36
Description: Hb response during weeks 28-36, was defined as mean Hb from 10-12 g/dL without receiving rescue therapy in the 6 weeks prior to, or during, the evaluation period. The percentages and 95% CI were unadjusted, the exact method of Clopper-Pearson was used for 95% CI. The Efficacy Emergent Period was defined as the evaluation period from the Analysis date of first dose intake up to end of treatment (EOT) Visit or last non-missing Hb assessment (for participants who died during the treatment period).
Time Frame: Weeks 28 to 36
Population: The analysis population was the PPS.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Roxadustat | ESA (Erythropoiesis-Stimulating Agent)
Number analyzed (Participants) | 386 | 397
Percentage of participants | 84.2 [80.2 to 87.7] | 82.4 [78.3 to 86.0]
Statistical Analysis 1: Comparison: Roxadustat vs ESA (Erythropoiesis-Stimulating Agent); A generalized linear model was used to estimate the difference in response rates between the arms, as an approximation for the Miettinen and Nurminen method, adjusting for following covariates: region, previous ESA treatment, cardiovascular history and baseline Hb as categorical variables; Test type: Non-Inferiority — Non-inferiority of roxadustat versus ESA (the non-inferiority margin for the difference between groups is -15%); p < 0.05, Miettinen and Nurminen — p-value for non-inferiority test based on 1-sided significance level; Difference of Percentages = 2.3, 95% CI 2-sided [-2.9 to 7.6]

4. Secondary Outcome: Change From BL in Low Density Lipoprotein Cholesterol (LDL-C) to the Average LDL-C of Weeks 12 to 28
Description: Baseline LDL was defined as the LDL value on Day 1. If this value was missing, the latest value prior to first study drug administration was used.
Time Frame: Baseline and weeks 12 to 28
Population: The analysis population was the FAS, with participants who had available data.
Measure: Least Squares Mean (95% Confidence Interval); unit: mmol/L
Arm/Group | Roxadustat | ESA (Erythropoiesis-Stimulating Agent)
Number analyzed (Participants) | 394 | 412
mmol/L | -0.459 [-0.517 to -0.401] | -0.082 [-0.138 to -0.026]
Statistical Analysis 1: Comparison: Roxadustat vs ESA (Erythropoiesis-Stimulating Agent); The model includes treatment arm, region, CV History, previous ESA treatment, visits and visit by treatment as categorical variables and baseline LDL, baseline Hb as continuous variables; Test type: Superiority; p < 0.001, Mixed Models Analysis — p-value for superiority test based on 2-sided significance level; LSM Difference = -0.377, 95% CI 2-sided [-0.451 to -0.304]

5. Secondary Outcome: Mean Monthly Intravenous (IV) Iron Use
Description: Participants with no or missing medication records of IV Iron have their monthly IV Iron use set to 0 mg. For participants who took IV Iron, but without a dosing frequency, the average values were set to missing.
Time Frame: Day 1 to week 36
Population: The analysis population was the FAS, with participants who had available data.
Measure: Least Squares Mean (95% Confidence Interval); unit: mg per month
Arm/Group | Roxadustat | ESA (Erythropoiesis-Stimulating Agent)
Number analyzed (Participants) | 413 | 419
mg per month | 21.6 [14.0 to 29.3] | 53.5 [46.0 to 61.1]
Statistical Analysis 1: Comparison: Roxadustat vs ESA (Erythropoiesis-Stimulating Agent); The model includes treatment arm, region, CV History, previous ESA treatment as categorical variables and baseline Hb as continuous variable; Test type: Superiority; p < 0.001, ANCOVA — p-value for superiority test based on 2-sided significance level; LSM Difference = -31.9, 95% CI 2-sided [-41.4 to -22.4]

6. Secondary Outcome: Change From BL in Short Form-36 (SF-36) Health Survey Physical Functioning (PF) Sub-score to the Average of Weeks 12 to 28
Description: Baseline SF-36 PF was defined as the SF-36 PF value on Day 1.The SF-36 is a Quality of Life (QoL) instrument designed to assess generic health concepts relevant across age, disease, and treatment groups. The SF-36 contains 36 items that measure eight scales: (1) physical functioning (PF); (2) role limitations due to physical health problems (RP); (3) bodily pain (BP); (4) social functioning (SF); (5) general health perceptions (GH); (6) role limitations due to emotional problems (RE); (7) vitality, energy or fatigue (VT); and (8) mental health(MH). Each scale is transformed into 0-100 score, with higher scores indicating better health status. The SF-36 PF consists of 11 questions focused on health and ability to do usual activities, with higher scores indicating better health status.
Time Frame: Baseline and weeks 12 to 28
Population: The analysis population was the PPS, with participants who had available data.
Measure: Least Squares Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | Roxadustat | ESA (Erythropoiesis-Stimulating Agent)
Number analyzed (Participants) | 376 | 391
Units on a scale | 0.050 [-0.640 to 0.740] | -0.155 [-0.825 to 0.514]
Statistical Analysis 1: Comparison: Roxadustat vs ESA (Erythropoiesis-Stimulating Agent); The model includes treatment arm, region, CV History, previous ESA treatment, visits (week 8, week 12, week 28) and visit by treatment as categorical variables, and baseline SF-36 PF, baseline Hb as continuous variables; Test type: Non-Inferiority — The margin for non-inferiority was -3; p < 0.05, Mixed Models Analysis — p-value for non-inferiority test based on 1-sided significance level; LSM Difference = 0.205, 95% CI 2-sided [-0.649 to 1.059]

7. Secondary Outcome: Change From BL in SF-36 Vitality (VT) Sub-score to the Average of Weeks 12 to 28
Description: Baseline VT Subscore was defined as the VT value on Day 1. The SF-36 is a QoL instrument designed to assess generic health concepts relevant across age, disease, and treatment groups. The SF-36 vitality has four questions with score range from 0-100 with higher scores indicating better vitality status.
Time Frame: Baseline and weeks 12 to 28
Population: The analysis population was the PPS, with participants who had available data.
Measure: Least Squares Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | Roxadustat | ESA (Erythropoiesis-Stimulating Agent)
Number analyzed (Participants) | 377 | 391
Units on a scale | 0.460 [-0.329 to 1.249] | -0.396 [-1.165 to 0.373]
Statistical Analysis 1: Comparison: Roxadustat vs ESA (Erythropoiesis-Stimulating Agent); The model includes treatment arm, region, CV History, previous ESA treatment, visits (week 8, week 12, week 28) and visit by treatment as categorical variables, and baseline SF-36 VT, baseline Hb as continuous variables; Test type: Non-Inferiority — The margin for non-inferiority was -3; p < 0.05, Mixed Models Analysis; LSM Difference = 0.856, 95% CI 2-sided [-0.115 to 1.828]

8. Secondary Outcome: Change From BL in Mean Arterial Pressure (MAP) to the Average of Weeks 20 to 28
Description: Baseline MAP was defined as the MAP value on Day 1. If this value was missing, the latest value prior to first study drug administration was used. Mean Arterial Pressure (MAP) is derived as: MAP = (2/3)*DBP + (1/3)*SBP.
Time Frame: Baseline and weeks 20 to 28
Population: The analysis population was the PPS, with participants who had available data.
Measure: Least Squares Mean (95% Confidence Interval); unit: mmHg
Arm/Group | Roxadustat | ESA (Erythropoiesis-Stimulating Agent)
Number analyzed (Participants) | 373 | 388
mmHg | -0.969 [-1.838 to -0.099] | -0.120 [-0.972 to 0.732]
Statistical Analysis 1: Comparison: Roxadustat vs ESA (Erythropoiesis-Stimulating Agent); The model includes treatment arm, region, CV History, previous ESA treatment, visits and visit by treatment as categorical variables, and baseline MAP, baseline Hb as continuous variables; Test type: Non-Inferiority — The margin for non-inferiority was 1; p < 0.05, Mixed Models Analysis — p-value for non-inferiority test based on 1-sided significance level; LSM Difference = -0.849, 95% CI 2-sided [-1.971 to 0.273]

9. Secondary Outcome: Time to First Occurrence of an Increase in Blood Pressure
Description: Increase in Blood Pressure was defined as either: Systolic Blood Pressure (SBP) ≥ 170 mmHg and an increase from BL ≥ 20 mmHg, or as: Diastolic Blood Pressure (DBP) ≥ 100 mmHg and an increase from BL ≥ 15 mmHg. For participants who have experienced more than one event, only their first event following study treatment was used. Data reported was analyzed by Kaplan-Meier estimate for cumulative proportion and the 95% confidence interval was calculated with Greenwood's formula.
Time Frame: Weeks 1 to 36
Population: The analysis population was the PPS, with participants who had available data.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- Roxadustat: Participants received roxadustat three times a week (TIW) for at least 52 weeks up to a maximum of 104 weeks. Participants received initial dose of roxadustat in doses of 100 mg, 150 mg or 200 mg, according to the average weekly dose of epoetin or darbepoetin alfa prior to randomization. Participants' roxadustat dosage was adjusted every 4 weeks to maintain Hb level within the target range 10.0 to 12.0 g/dL. Dose adjustment steps were as follows: 20, 40, 50, 70, 100, 150, 200, 250, 300, and 400 mg. Oral iron treatment of 200 mg was allowed for supplementation to support erythropoiesis. Treatment with intravenous iron was allowed only if certain protocol criteria were met. .
Arm/Group | Roxadustat | ESA (Erythropoiesis-Stimulating Agent)
Number analyzed (Participants) | 386 | 397
Percentage of participants
  Week 12 | 11.7 [8.5 to 14.9] | 11.1 [8.0 to 14.2]
  Week 24 | 15.9 [12.2 to 19.6] | 15.4 [11.9 to 19.0]
  Week 36 | 21.1 [14.0 to 28.2] | 23.5 [16. to 30.9]
Statistical Analysis 1: Comparison: Roxadustat vs ESA (Erythropoiesis-Stimulating Agent); Hazard Ratio was calculated using stratified Cox Proportional Hazards regression stratifying on region, CV history, previous ESA treatment, and adjusting on Hb at baseline as continuous covariate. Non-inferiority was declared if the upper bound of the 95% CI is below 1.3; Test type: Non-Inferiority — Non-inferiority (hazard ratio margin of 1.3); p < 0.05, Regression, Cox — p-value for non-inferiority test based on 1-sided significance level; Hazard Ratio (HR) = 0.924, 95% CI 2-sided [0.669 to 1.276]

10. Secondary Outcome: Change From BL in Mean Arterial Pressure (MAP) to the Average MAP Value of Weeks 20 to 28
Description: as for outcome 8
Time Frame: Baseline and weeks 20 to 28
Population: The analysis population was the FAS, with participants who had available data.
Measure: Least Squares Mean (95% Confidence Interval); unit: mmHg
Arm/Group | Roxadustat | ESA (Erythropoiesis-Stimulating Agent)
Number analyzed (Participants) | 381 | 401
mmHg | -0.739 [-1.600 to 0.123] | -0.160 [-0.997 to 0.678]
Statistical Analysis 1: Comparison: Roxadustat vs ESA (Erythropoiesis-Stimulating Agent); [analysis description as in outcome 8, analysis 1]; Test type: Superiority; p = 0.308, Mixed Models Analysis — p-value for superiority test based on 2-sided significance level; LSM Difference = -0.579, 95% CI 2-sided [-1.694 to 0.536]

11. Secondary Outcome: Time to First Occurrence of an Increase in Blood Pressure
Description: Increase in Blood Pressure was defined as either: SBP ≥ 170 mmHg and an increase from BL ≥ 20 mmHg, or as: DBP ≥ 100 mmHg and an increase from BL ≥ 15 mmHg. Data reported was analyzed by Kaplan-Meier estimate for cumulative proportion and the 95% confidence interval was calculated with Greenwood's formula.
Time Frame: Weeks 1 to 36
Population: The analysis population was the FAS, with participants who had available data.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Roxadustat | ESA (Erythropoiesis-Stimulating Agent)
Number analyzed (Participants) | 413 | 420
Percentage of participants
  Week 12 | 11.6 [8.5 to 14.8] | 12.0 [8.9 to 15.1]
  Week 24 | 16.1 [12.5 to 19.7] | 16.2 [12.6 to 19.7]
  Week 36 | 21.2 [14.1 to 28.3] | 24.1 [16.7 to 31.4]
Statistical Analysis 1: Comparison: Roxadustat vs ESA (Erythropoiesis-Stimulating Agent); Hazard Ratio was calculated using stratified Cox Proportional Hazards regression stratifying on region, CV history, previous ESA treatment, and adjusting on Hb at baseline as continuous covariate. Superiority was declared if the upper bound of the 95% CI is lower than 1; Test type: Superiority; p = 0.582, Regression, Cox — p-value for superiority test based on 2-sided significance level; Hazard Ratio (HR) = 0.915, 95% CI 2-sided [0.668 to 1.254]

12. Secondary Outcome: Percentage of Participants With a Hb Response During Weeks 28 and 36 Regardless of Use of Rescue Therapy
Description: Hb response was defined as mean Hb during weeks 28 to 36 within the target range of 10.0 to 12.0 g/dL. The percentages and 95% CI are unadjusted, the exact method of Clopper-Pearson was used for 95% CI.
Time Frame: Weeks 28 to 36
Population: The analysis population was the FAS.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Roxadustat | ESA (Erythropoiesis-Stimulating Agent)
Number analyzed (Participants) | 413 | 420
Percentage of participants | 83.1 [79.1 to 86.5] | 82.1 [78.1 to 85.7]
Statistical Analysis 1: Comparison: Roxadustat vs ESA (Erythropoiesis-Stimulating Agent); [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.609, Miettinen and Nurminen method — p-value for superiority test based on 2-sided significance level; Difference of Percentages = 1.4, 95% CI 2-sided [-3.8 to 6.5]

13. Secondary Outcome: Change From BL in Hb to Each Postdosing Time Point
Description: Baseline Hb was defined as the mean of four latest central laboratory Hb values prior or on the same date as first study drug intake (pre-dose).
Time Frame: Baseline and weeks 1, 2, 3, 4, 5, 6, 7, 8, 10, 12, 14, 16, 18,20, 22, 24, 26, 28, 30, 32, 34, 36, 40, 44, 48, 52, 56, 60, 64, 68, 72,76, 80, 84, 88, 92, 96, 100, and 104
Population: The analysis population was the FAS.
Measure: Least Squares Mean (95% Confidence Interval); unit: g/dL
Arm/Group | Roxadustat | ESA (Erythropoiesis-Stimulating Agent)
Number analyzed (Participants) | 413 | 420
g/dL
  Hb Change From BL to Week 1: number analyzed (Participants) | 407 | 411
  Hb Change From BL to Week 1 | 0.232 [0.164 to 0.300] | 0.068 [0.000 to 0.135]
  Hb Change From BL to Week 2: number analyzed (Participants) | 401 | 411
  Hb Change From BL to Week 2 | 0.496 [0.420 to 0.572] | 0.054 [-0.022 to 0.129]
  Hb Change From BL to Week 3: number analyzed (Participants) | 394 | 408
  Hb Change From BL to Week 3 | 0.633 [0.552 to 0.714] | 0.071 [-0.008 to 0.151]
  Hb Change From BL to Week 4: number analyzed (Participants) | 399 | 413
  Hb Change From BL to Week 4 | 0.803 [0.715 to 0.891] | 0.095 [0.009 to 0.181]
  Hb Change From BL to Week 5: number analyzed (Participants) | 399 | 407
  Hb Change From BL to Week 5 | 0.723 [0.633 to 0.812] | -0.045 [-0.133 to 0.043]
  Hb Change From BL to Week 6: number analyzed (Participants) | 391 | 405
  Hb Change From BL to Week 6 | 0.868 [0.776 to 0.959] | 0.138 [0.048 to 0.228]
  Hb Change From BL to Week 7: number analyzed (Participants) | 389 | 404
  Hb Change From BL to Week 7 | 0.698 [0.606 to 0.791] | -0.031 [-0.122 to 0.060]
  Hb Change From BL to Week 8: number analyzed (Participants) | 393 | 402
  Hb Change From BL to Week 8 | 0.816 [0.724 to 0.907] | 0.116 [0.026 to 0.206]
  Hb Change From BL to Week 10: number analyzed (Participants) | 396 | 409
  Hb Change From BL to Week 10 | 0.640 [0.546 to 0.735] | -0.019 [-0.111 to 0.073]
  Hb Change From BL to Week 12: number analyzed (Participants) | 384 | 399
  Hb Change From BL to Week 12 | 0.732 [0.634 to 0.830] | 0.139 [0.043 to 0.235]
  Hb Change From BL to Week 14: number analyzed (Participants) | 383 | 400
  Hb Change From BL to Week 14 | 0.508 [0.408 to 0.608] | 0.005 [-0.093 to 0.103]
  Hb Change From BL to Week 16: number analyzed (Participants) | 381 | 401
  Hb Change From BL to Week 16 | 0.613 [0.511 to 0.716] | 0.244 [0.144 to 0.344]
  Hb Change From BL to Week 18: number analyzed (Participants) | 378 | 395
  Hb Change From BL to Week 18 | 0.380 [0.283 to 0.477] | 0.017 [-0.078 to 0.112]
  Hb Change From BL to Week 20: number analyzed (Participants) | 376 | 394
  Hb Change From BL to Week 20 | 0.501 [0.405 to 0.596] | 0.217 [0.124 to 0.309]
  Hb Change From BL to Week 22: number analyzed (Participants) | 370 | 395
  Hb Change From BL to Week 22 | 0.266 [0.170 to 0.363] | 0.069 [-0.025 to 0.163]
  Hb Change From BL to Week 24: number analyzed (Participants) | 362 | 388
  Hb Change From BL to Week 24 | 0.262 [0.168 to 0.356] | 0.075 [-0.017 to 0.166]
  Hb Change From BL to Week 26: number analyzed (Participants) | 359 | 387
  Hb Change From BL to Week 26 | 0.316 [0.220 to 0.412] | 0.073 [-0.020 to 0.165]
  Hb Change From BL to Week 28: number analyzed (Participants) | 360 | 388
  Hb Change From BL to Week 28 | 0.549 [0.452 to 0.647] | 0.342 [0.248 to 0.437]
  Hb Change From BL to Week 30: number analyzed (Participants) | 352 | 380
  Hb Change From BL to Week 30 | 0.333 [0.236 to 0.429] | 0.106 [0.013 to 0.198]
  Hb Change From BL to Week 32: number analyzed (Participants) | 346 | 376
  Hb Change From BL to Week 32 | 0.310 [0.211 to 0.409] | 0.111 [0.016 to 0.207]
  Hb Change From BL to Week 34: number analyzed (Participants) | 342 | 374
  Hb Change From BL to Week 34 | 0.364 [0.268 to 0.460] | 0.084 [-0.007 to 0.176]
  Hb Change From BL to Week 36: number analyzed (Participants) | 339 | 373
  Hb Change From BL to Week 36 | 0.482 [0.382 to 0.581] | 0.225 [0.130 to 0.320]
  Hb Change From BL to Week 40: number analyzed (Participants) | 336 | 373
  Hb Change From BL to Week 40 | 0.199 [0.095 to 0.304] | 0.064 [-0.036 to 0.163]
  Hb Change From BL to Week 44: number analyzed (Participants) | 328 | 367
  Hb Change From BL to Week 44 | 0.335 [0.221 to 0.448] | 0.252 [0.145 to 0.360]
  Hb Change From BL to Week 48: number analyzed (Participants) | 323 | 365
  Hb Change From BL to Week 48 | 0.158 [0.047 to 0.270] | 0.131 [0.027 to 0.236]
  Hb Change From BL to Week 52: number analyzed (Participants) | 308 | 363
  Hb Change From BL to Week 52 | 0.385 [0.273 to 0.496] | 0.186 [0.082 to 0.290]
  Hb Change From BL to Week 56: number analyzed (Participants) | 311 | 360
  Hb Change From BL to Week 56 | 0.217 [0.104 to 0.329] | 0.069 [-0.035 to 0.174]
  Hb Change From BL to Week 60: number analyzed (Participants) | 299 | 353
  Hb Change From BL to Week 60 | 0.368 [0.256 to 0.479] | 0.171 [0.067 to 0.275]
  Hb Change From BL to Week 64: number analyzed (Participants) | 289 | 344
  Hb Change From BL to Week 64 | 0.181 [0.067 to 0.295] | -0.093 [-0.198 to 0.012]
  Hb Change From BL to Week 68: number analyzed (Participants) | 290 | 349
  Hb Change From BL to Week 68 | 0.306 [0.195 to 0.416] | 0.100 [-0.002 to 0.202]
  Hb Change From BL to Week 72: number analyzed (Participants) | 284 | 339
  Hb Change From BL to Week 72 | 0.109 [-0.005 to 0.222] | -0.009 [-0.113 to 0.095]
  Hb Change From BL to Week 76: number analyzed (Participants) | 278 | 338
  Hb Change From BL to Week 76 | 0.401 [0.280 to 0.521] | 0.189 [0.079 to 0.299]
  Hb Change From BL to Week 80: number analyzed (Participants) | 274 | 327
  Hb Change From BL to Week 80 | 0.087 [-0.028 to 0.203] | -0.015 [-0.120 to 0.091]
  Hb Change From BL to Week 84: number analyzed (Participants) | 270 | 328
  Hb Change From BL to Week 84 | 0.318 [0.199 to 0.438] | 0.126 [0.017 to 0.235]
  Hb Change From BL to Week 88: number analyzed (Participants) | 258 | 326
  Hb Change From BL to Week 88 | 0.026 [-0.091 to 0.144] | -0.018 [-0.124 to 0.088]
  Hb Change From BL to Week 92: number analyzed (Participants) | 255 | 313
  Hb Change From BL to Week 92 | 0.357 [0.232 to 0.483] | 0.154 [0.041 to 0.267]
  Hb Change From BL to Week 96: number analyzed (Participants) | 253 | 312
  Hb Change From BL to Week 96 | 0.126 [0.010 to 0.242] | -0.058 [-0.163 to 0.046]
  Hb Change From BL to Week 100: number analyzed (Participants) | 248 | 311
  Hb Change From BL to Week 100 | 0.302 [0.175 to 0.430] | 0.138 [0.024 to 0.253]
  Hb Change From BL to Week 104: number analyzed (Participants) | 240 | 299
  Hb Change From BL to Week 104 | 0.232 [0.100 to 0.363] | 0.133 [0.014 to 0.251]
Statistical Analysis 1: Comparison: Roxadustat vs ESA (Erythropoiesis-Stimulating Agent); Week 1- The model included treatment, visit, visit by treatment interaction, Previous ESA Treatment, region and history of CV disease as fixed class factors and baseline Hb as continuous covariates; Test type: Superiority; p < 0.001, Mixed Models Analysis — p-value for superiority test based on 2-sided significance level; LSM Difference = 0.164, 95% CI 2-sided [0.072 to 0.256]
Statistical Analysis 2: Comparison: Roxadustat vs ESA (Erythropoiesis-Stimulating Agent); Week 2- The model included treatment, visit, visit by treatment interaction, Previous ESA Treatment, region and history of CV disease as fixed class factors and baseline Hb as continuous covariates; Test type: Superiority; p < 0.001, Mixed Models Analysis — p-value for superiority test based on 2-sided significance level; LSM Difference = 0.443, 95% CI 2-sided [0.339 to 0.546]
Statistical Analysis 3: Comparison: Roxadustat vs ESA (Erythropoiesis-Stimulating Agent); Week 3 - The model included treatment, visit, visit by treatment interaction, Previous ESA Treatment, region and history of CV disease as fixed class factors and baseline Hb as continuous covariates; Test type: Superiority; p < 0.001, Mixed Models Analysis — p-value for superiority test based on 2-sided significance level; LSM Difference = 0.561, 95% CI 2-sided [0.451 to 0.672]
Statistical Analysis 4: Comparison: Roxadustat vs ESA (Erythropoiesis-Stimulating Agent); Week 4 - The model included treatment, visit, visit by treatment interaction, Previous ESA Treatment, region and history of CV disease as fixed class factors and baseline Hb as continuous covariates; Test type: Superiority; p < 0.001, Mixed Models Analysis — p-value for superiority test based on 2-sided significance level; LSM Difference = 0.708, 95% CI [0.588 to 0.828]
Statistical Analysis 5: Comparison: Roxadustat vs ESA (Erythropoiesis-Stimulating Agent); Week 5 - The model included treatment, visit, visit by treatment interaction, Previous ESA Treatment, region and history of CV disease as fixed class factors and baseline Hb as continuous covariates; Test type: Superiority; p < 0.001, Mixed Models Analysis — p-value for superiority test based on 2-sided significance level; LSM Difference = 0.768, 95% CI 2-sided [0.645 to 0.890]
Statistical Analysis 6: Comparison: Roxadustat vs ESA (Erythropoiesis-Stimulating Agent); Week 6 - The model included treatment, visit, visit by treatment interaction, Previous ESA Treatment, region and history of CV disease as fixed class factors and baseline Hb as continuous covariates; Test type: Superiority; p < 0.001, Mixed Models Analysis — p-value for superiority test based on 2-sided significance level; LSM Difference = 0.729, 95% CI 2-sided [0.604 to 0.855]
Statistical Analysis 7: Comparison: Roxadustat vs ESA (Erythropoiesis-Stimulating Agent); Week 7 - The model included treatment, visit, visit by treatment interaction, Previous ESA Treatment, region and history of CV disease as fixed class factors and baseline Hb as continuous covariates; Test type: Superiority; p < 0.001, Mixed Models Analysis — p-value for superiority test based on 2-sided significance level; LSM Difference = 0.729, 95% CI 2-sided [0.603 to 0.856]
Statistical Analysis 8: Comparison: Roxadustat vs ESA (Erythropoiesis-Stimulating Agent); Week 8 - The model included treatment, visit, visit by treatment interaction, Previous ESA Treatment, region and history of CV disease as fixed class factors and baseline Hb as continuous covariates; Test type: Superiority; p < 0.001, Mixed Models Analysis — p-value for superiority test based on 2-sided significance level; LSM Difference = 0.700, 95% CI 2-sided [0.574 to 0.826]
Statistical Analysis 9: Comparison: Roxadustat vs ESA (Erythropoiesis-Stimulating Agent); Week 10 - The model included treatment, visit, visit by treatment interaction, Previous ESA Treatment, region and history of CV disease as fixed class factors and baseline Hb as continuous covariates; Test type: Superiority; p < 0.001, Mixed Models Analysis — p-value for superiority test based on 2-sided significance level; LSM Difference = 0.659, 95% CI 2-sided [0.530 to 0.788]
Statistical Analysis 10: Comparison: Roxadustat vs ESA (Erythropoiesis-Stimulating Agent); Week 12 - The model included treatment, visit, visit by treatment interaction, Previous ESA Treatment, region and history of CV disease as fixed class factors and baseline Hb as continuous covariates; Test type: Superiority; p < 0.001, Mixed Models Analysis — p-value for superiority test based on 2-sided significance level; LSM Difference = 0.593, 95% CI 2-sided [0.459 to 0.727]
Statistical Analysis 11: Comparison: Roxadustat vs ESA (Erythropoiesis-Stimulating Agent); Week 14 - The model included treatment, visit, visit by treatment interaction, Previous ESA Treatment, region and history of CV disease as fixed class factors and baseline Hb as continuous covariates; Test type: Superiority; p < 0.001, Mixed Models Analysis — p-value for superiority test based on 2-sided significance level; LSM Difference = 0.503, 95% CI 2-sided [0.366 to 0.640]
Statistical Analysis 12: Comparison: Roxadustat vs ESA (Erythropoiesis-Stimulating Agent); Week 16 - The model included treatment, visit, visit by treatment interaction, Previous ESA Treatment, region and history of CV disease as fixed class factors and baseline Hb as continuous covariates; Test type: Superiority; p < 0.001, Mixed Models Analysis — p-value for superiority test based on 2-sided significance level; LSM Difference = 0.369, 95% CI 2-sided [0.229 to 0.510]
Statistical Analysis 13: Comparison: Roxadustat vs ESA (Erythropoiesis-Stimulating Agent); Week 18 - The model included treatment, visit, visit by treatment interaction, Previous ESA Treatment, region and history of CV disease as fixed class factors and baseline Hb as continuous covariates; Test type: Superiority; p < 0.001, Mixed Models Analysis — p-value for superiority test based on 2-sided significance level; LSM Difference = 0.363, 95% CI 2-sided [0.230 to 0.496]
Statistical Analysis 14: Comparison: Roxadustat vs ESA (Erythropoiesis-Stimulating Agent); Week 20 - The model included treatment, visit, visit by treatment interaction, Previous ESA Treatment, region and history of CV disease as fixed class factors and baseline Hb as continuous covariates; Test type: Superiority; p < 0.001, Mixed Models Analysis — p-value for superiority test based on 2-sided significance level; LSM Difference = 0.284, 95% CI 2-sided [0.154 to 0.414]
Statistical Analysis 15: Comparison: Roxadustat vs ESA (Erythropoiesis-Stimulating Agent); Week 22 - The model included treatment, visit, visit by treatment interaction, Previous ESA Treatment, region and history of CV disease as fixed class factors and baseline Hb as continuous covariates; Test type: Superiority; p = 0.003, Mixed Models Analysis — p-value for superiority test based on 2-sided significance level; LSM Difference = 0.197, 95% CI 2-sided [0.065 to 0.329]
Statistical Analysis 16: Comparison: Roxadustat vs ESA (Erythropoiesis-Stimulating Agent); Week 24 - The model included treatment, visit, visit by treatment interaction, Previous ESA Treatment, region and history of CV disease as fixed class factors and baseline Hb as continuous covariates; Test type: Superiority; p = 0.004, Mixed Models Analysis — p-value for superiority test based on 2-sided significance level; LSM Difference = 0.187, 95% CI 2-sided [0.059 to 0.316]
Statistical Analysis 17: Comparison: Roxadustat vs ESA (Erythropoiesis-Stimulating Agent); Week 26 - The model included treatment, visit, visit by treatment interaction, Previous ESA Treatment, region and history of CV disease as fixed class factors and baseline Hb as continuous covariates; Test type: Superiority; p < 0.001, Mixed Models Analysis — p-value for superiority test based on 2-sided significance level; LSM Difference = 0.243, 95% CI 2-sided [0.113 to 0.373]
Statistical Analysis 18: Comparison: Roxadustat vs ESA (Erythropoiesis-Stimulating Agent); Week 28 - The model included treatment, visit, visit by treatment interaction, Previous ESA Treatment, region and history of CV disease as fixed class factors and baseline Hb as continuous covariates; Test type: Superiority; p = 0.002, Mixed Models Analysis — p-value for superiority test based on 2-sided significance level; LSM Difference = 0.207, 95% CI 2-sided [0.074 to 0.340]
Statistical Analysis 19: Comparison: Roxadustat vs ESA (Erythropoiesis-Stimulating Agent); Week 30 - The model included treatment, visit, visit by treatment interaction, Previous ESA Treatment, region and history of CV disease as fixed class factors and baseline Hb as continuous covariates; Test type: Superiority; p < 0.001, Mixed Models Analysis — p-value for superiority test based on 2-sided significance level; LSM Difference = 0.227, 95% CI 2-sided [0.096 to 0.358]
Statistical Analysis 20: Comparison: Roxadustat vs ESA (Erythropoiesis-Stimulating Agent); Week 32 - The model included treatment, visit, visit by treatment interaction, Previous ESA Treatment, region and history of CV disease as fixed class factors and baseline Hb as continuous covariates; Test type: Superiority; p = 0.004, Mixed Models Analysis; p-value for superiority test based on 2-sided significance level; LSM Difference = 0.199, 95% CI 2-sided [0.064 to 0.334]
Statistical Analysis 21: Comparison: Roxadustat vs ESA (Erythropoiesis-Stimulating Agent); Week 34 - The model included treatment, visit, visit by treatment interaction, Previous ESA Treatment, region and history of CV disease as fixed class factors and baseline Hb as continuous covariates; Test type: Superiority; p < 0.001, Mixed Models Analysis — p-value for superiority test based on 2-sided significance level; LSM Difference = 0.279, 95% CI [0.150 to 0.409]
Statistical Analysis 22: Comparison: Roxadustat vs ESA (Erythropoiesis-Stimulating Agent); Week 36- The model included treatment, visit, visit by treatment interaction, Previous ESA Treatment, region and history of CV disease as fixed class factors and baseline Hb as continuous covariates; Test type: Superiority; p < 0.001, Mixed Models Analysis — p-value for superiority test based on 2-sided significance level; LSM Difference = 0.256, 95% CI 2-sided [0.121 to 0.391]
Statistical Analysis 23: Comparison: Roxadustat vs ESA (Erythropoiesis-Stimulating Agent); Week 40 - The model included treatment, visit, visit by treatment interaction, Previous ESA Treatment, region and history of CV disease as fixed class factors and baseline Hb as continuous covariates; Test type: Superiority; p = 0.060, Mixed Models Analysis — p-value for superiority test based on 2-sided significance level; LSM Difference = 0.136, 95% CI 2-sided [-0.006 to 0.277]
Statistical Analysis 24: Comparison: Roxadustat vs ESA (Erythropoiesis-Stimulating Agent); Week 44 - The model included treatment, visit, visit by treatment interaction, Previous ESA Treatment, region and history of CV disease as fixed class factors and baseline Hb as continuous covariates; Test type: Superiority; p = 0.293, Mixed Models Analysis — p-value for superiority test based on 2-sided significance level; LSM Difference = 0.082, 95% CI 2-sided [-0.071 to 0.236]
Statistical Analysis 25: Comparison: Roxadustat vs ESA (Erythropoiesis-Stimulating Agent); Week 48 - The model included treatment, visit, visit by treatment interaction, Previous ESA Treatment, region and history of CV disease as fixed class factors and baseline Hb as continuous covariates; Test type: Superiority; p = 0.723, Mixed Models Analysis — p-value for superiority test based on 2-sided significance level; LSM Difference = 0.027, 95% CI 2-sided [-0.123 to 0.177]
Statistical Analysis 26: Comparison: Roxadustat vs ESA (Erythropoiesis-Stimulating Agent); Week 52 - The model included treatment, visit, visit by treatment interaction, Previous ESA Treatment, region and history of CV disease as fixed class factors and baseline Hb as continuous covariates; Test type: Superiority; p = 0.009, Mixed Models Analysis — p-value for superiority test based on 2-sided significance level; LSM Difference = 0.199, 95% CI 2-sided [0.049 to 0.348]
Statistical Analysis 27: Comparison: Roxadustat vs ESA (Erythropoiesis-Stimulating Agent); Week 56 - The model included treatment, visit, visit by treatment interaction, Previous ESA Treatment, region and history of CV disease as fixed class factors and baseline Hb as continuous covariates; Test type: Superiority; p = 0.056, Mixed Models Analysis — p-value for superiority test based on 2-sided significance level; LSM Difference = 0.147, 95% CI 2-sided [-0.004 to 0.298]
Statistical Analysis 28: Comparison: Roxadustat vs ESA (Erythropoiesis-Stimulating Agent); Week 60 - The model included treatment, visit, visit by treatment interaction, Previous ESA Treatment, region and history of CV disease as fixed class factors and baseline Hb as continuous covariates; Test type: Superiority; p = 0.010, Mixed Models Analysis — p-value for superiority test based on 2-sided significance level; LSM Difference = 0.196, 95% CI 2-sided [0.047 to 0.346]
Statistical Analysis 29: Comparison: Roxadustat vs ESA (Erythropoiesis-Stimulating Agent); Week 64 - The model included treatment, visit, visit by treatment interaction, Previous ESA Treatment, region and history of CV disease as fixed class factors and baseline Hb as continuous covariates; Test type: Superiority; p < 0.001, Mixed Models Analysis — p-value for superiority test based on 2-sided significance level; LSM Difference = 0.275, 95% CI 2-sided [0.123 to 0.427]
Statistical Analysis 30: Comparison: Roxadustat vs ESA (Erythropoiesis-Stimulating Agent); Week 68 - The model included treatment, visit, visit by treatment interaction, Previous ESA Treatment, region and history of CV disease as fixed class factors and baseline Hb as continuous covariates; Test type: Superiority; p = 0.006, Mixed Models Analysis — p-value for superiority test based on 2-sided significance level; LSM Difference = 0.206, 95% CI 2-sided [0.059 to 0.353]
Statistical Analysis 31: Comparison: Roxadustat vs ESA (Erythropoiesis-Stimulating Agent); Week 72 - The model included treatment, visit, visit by treatment interaction, Previous ESA Treatment, region and history of CV disease as fixed class factors and baseline Hb as continuous covariates; Test type: Superiority; p = 0.127, Mixed Models Analysis — p-value for superiority test based on 2-sided significance level; LSM Difference = 0.118, 95% CI 2-sided [-0.033 to 0.269]
Statistical Analysis 32: Comparison: Roxadustat vs ESA (Erythropoiesis-Stimulating Agent); Week 76 - The model included treatment, visit, visit by treatment interaction, Previous ESA Treatment, region and history of CV disease as fixed class factors and baseline Hb as continuous covariates; Test type: Superiority; p = 0.010, Mixed Models Analysis — p-value for superiority test based on 2-sided significance level; LSM Difference = 0.211, 95% CI 2-sided [0.051 to 0.371]
Statistical Analysis 33: Comparison: Roxadustat vs ESA (Erythropoiesis-Stimulating Agent); Week 80 - The model included treatment, visit, visit by treatment interaction, Previous ESA Treatment, region and history of CV disease as fixed class factors and baseline Hb as continuous covariates; Test type: Superiority; p = 0.191, Mixed Models Analysis — p-value for superiority test based on 2-sided significance level; LSM Difference = 0.102, 95% CI 2-sided [-0.051 to 0.255]
Statistical Analysis 34: Comparison: Roxadustat vs ESA (Erythropoiesis-Stimulating Agent); Week 84 - The model included treatment, visit, visit by treatment interaction, Previous ESA Treatment, region and history of CV disease as fixed class factors and baseline Hb as continuous covariates; Test type: Superiority; p = 0.018, Mixed Models Analysis — p-value for superiority test based on 2-sided significance level; LSM Difference = 0.192, 95% CI 2-sided [0.033 to 0.351]
Statistical Analysis 35: Comparison: Roxadustat vs ESA (Erythropoiesis-Stimulating Agent); Week 88 - The model included treatment, visit, visit by treatment interaction, Previous ESA Treatment, region and history of CV disease as fixed class factors and baseline Hb as continuous covariates; Test type: Superiority; p = 0.576, Mixed Models Analysis — p-value for superiority test based on 2-sided significance level; LSM Difference = 0.044, 95% CI 2-sided [-0.111 to 0.200]
Statistical Analysis 36: Comparison: Roxadustat vs ESA (Erythropoiesis-Stimulating Agent); Week 92 - The model included treatment, visit, visit by treatment interaction, Previous ESA Treatment, region and history of CV disease as fixed class factors and baseline Hb as continuous covariates; Test type: Superiority; p = 0.017, Mixed Models Analysis — p-value for superiority test based on 2-sided significance level; LSM Difference = 0.203, 95% CI 2-sided [0.037 to 0.369]
Statistical Analysis 37: Comparison: Roxadustat vs ESA (Erythropoiesis-Stimulating Agent); Week 96 - The model included treatment, visit, visit by treatment interaction, Previous ESA Treatment, region and history of CV disease as fixed class factors and baseline Hb as continuous covariates; Test type: Superiority; p = 0.019, Mixed Models Analysis — p-value for superiority test based on 2-sided significance level; LSM Difference = 0.184, 95% CI 2-sided [0.031 to 0.338]
Statistical Analysis 38: Comparison: Roxadustat vs ESA (Erythropoiesis-Stimulating Agent); Week 100 - The model included treatment, visit, visit by treatment interaction, Previous ESA Treatment, region and history of CV disease as fixed class factors and baseline Hb as continuous covariates; Test type: Superiority; p = 0.056, Mixed Models Analysis — p-value for superiority test based on 2-sided significance level; LSM Difference = 0.164, 95% CI [-0.004 to 0.333]
Statistical Analysis 39: Comparison: Roxadustat vs ESA (Erythropoiesis-Stimulating Agent); Week 104 - The model included treatment, visit, visit by treatment interaction, Previous ESA Treatment, region and history of CV disease as fixed class factors and baseline Hb as continuous covariates; Test type: Superiority; p = 0.267, Mixed Models Analysis — p-value for superiority test based on 2-sided significance level; LSM Difference = 0.099, 95% CI 2-sided [-0.076 to 0.273]

14. Secondary Outcome: Hb Level Averaged Over Weeks 28 to 36, 44 to 52, and 96 to 104 Without Use of Rescue Therapy
Description: Baseline Hb was defined as the mean of four latest central laboratory Hb values prior or on the same date as first study drug intake (pre-dose). Averaged Hb values over weeks 28-36, weeks 44-52 and weeks 96-104 are observed values.
Time Frame: Weeks 28 to 36, 44 to 52, and 96 to 104
Population: The analysis population was the FAS.
Measure: Least Squares Mean (95% Confidence Interval); unit: g/dL
Arm/Group | Roxadustat | ESA (Erythropoiesis-Stimulating Agent)
Number analyzed (Participants) | 413 | 420
g/dL
  Average Hb Over Weeks 28-36: number analyzed (Participants) | 362 | 393
  Average Hb Over Weeks 28-36 | 11.183 [11.100 to 11.265] | 10.946 [10.867 to 11.025]
  Average Hb Over Weeks 44-52: number analyzed (Participants) | 330 | 370
  Average Hb Over Weeks 44-52 | 11.099 [11.009 to 11.189] | 10.994 [10.909 to 11.079]
  Average Hb Over Weeks 96-104: number analyzed (Participants) | 252 | 317
  Average Hb Over Weeks 96-104 | 11.007 [10.904 to 11.110] | 10.858 [10.766 to 10.950]
Statistical Analysis 1: Comparison: Roxadustat vs ESA (Erythropoiesis-Stimulating Agent); Weeks 28-36 - The model includes treatment arm, region, CV History, previous ESA treatment, visits and visit by treatment as categorical variables and baseline Hb as continuous variable; Test type: Superiority; p < 0.001, Mixed Models Analysis — p-value for superiority test based on 2-sided significance level; LSM Difference = 0.237, 95% CI 2-sided [0.127 to 0.347]
Statistical Analysis 2: Comparison: Roxadustat vs ESA (Erythropoiesis-Stimulating Agent); Weeks 44-52 - The model includes treatment arm, region, CV History, previous ESA treatment, visits and visit by treatment as categorical variables and baseline Hb as continuous variable; Test type: Superiority; p = 0.086, Mixed Models Analysis — p-value for superiority test based on 2-sided significance level; LSM Difference = 0.105, 95% CI 2-sided [-0.015 to 0.225]
Statistical Analysis 3: Comparison: Roxadustat vs ESA (Erythropoiesis-Stimulating Agent); Weeks 96-104 - The model includes treatment arm, region, CV History, previous ESA treatment, visits and visit by treatment as categorical variables and baseline Hb as continuous variable; Test type: Superiority; p = 0.031, Mixed Models Analysis — p-value for superiority test based on 2-sided significance level; LSM Difference = 0.149, 95% CI 2-sided [0.014 to 0.284]

15. Secondary Outcome: Change From BL in Hb to the Average of Weeks 28 to 36, 44 to 52, and 96 to 104 Regardless of the Use of Rescue Therapy
Description: Change from baseline to the average Hb are observed values. Baseline Hb was defined as the mean of four latest central laboratory Hb values prior or on the same date as first study drug intake (pre-dose).
Time Frame: Baseline and weeks 28 to 36, 44 to 52, and 96 to 104
Population: The analysis population was the FAS.
Measure: Least Squares Mean (95% Confidence Interval); unit: g/dL
Arm/Group | Roxadustat | ESA (Erythropoiesis-Stimulating Agent)
Number analyzed (Participants) | 413 | 420
g/dL
  Hb Change From BL to Weeks 28-36: number analyzed (Participants) | 364 | 393
  Hb Change From BL to Weeks 28-36 | 0.408 [0.325 to 0.491] | 0.173 [0.093 to 0.252]
  Hb Change From BL to Weeks 44-52: number analyzed (Participants) | 331 | 371
  Hb Change From BL to Weeks 44-52 | 0.298 [0.203 to 0.394] | 0.194 [0.104 to 0.284]
  Hb Change From BL to Weeks 96-104: number analyzed (Participants) | 254 | 318
  Hb Change From BL to Weeks 96-104 | 0.225 [0.119 to 0.331] | 0.076 [-0.020 to 0.171]
Statistical Analysis 1: Comparison: Roxadustat vs ESA (Erythropoiesis-Stimulating Agent); [analysis description as in outcome 14, analysis 1]; Test type: Superiority; p < 0.001, Mixed Models Analysis; LSM Difference = 0.235, 95% CI 2-sided [0.125 to 0.346]
Statistical Analysis 2: Comparison: Roxadustat vs ESA (Erythropoiesis-Stimulating Agent); [analysis description as in outcome 14, analysis 2]; Test type: Superiority; p = 0.110, Mixed Models Analysis; LSM Difference = 0.104, 95% CI 2-sided [-0.024 to 0.232]
Statistical Analysis 3: Comparison: Roxadustat vs ESA (Erythropoiesis-Stimulating Agent); [analysis description as in outcome 14, analysis 3]; Test type: Superiority; p = 0.036, Mixed Models Analysis; LSM Difference = 0.149, 95% CI 2-sided [0.010 to 0.288]

16. Secondary Outcome: Percentage of Hb Values ≥ 10 g/dL in Weeks 28 to 36, 44 to 52, and 96 to 104 Without Use of Rescue Therapy
Description: Percentage for each participant was calculated as Number of Hb values >= 10.0 g/dL / Total number of Hb values*100 in weeks 28 to 36, 44 to 52 and 96 to 104 without use of rescue therapy within 6 weeks prior to and during the 8 week evaluation period.
Time Frame: Weeks 28-36, 44-52 and 96-104
Population: The analysis population was the FAS.
Measure: Mean (Standard Deviation); unit: percentage of Hb values
Arm/Group | Roxadustat | ESA (Erythropoiesis-Stimulating Agent)
Number analyzed (Participants) | 413 | 420
percentage of Hb values
  Weeks 28-36: number analyzed (Participants) | 364 | 393
  Weeks 28-36 | 93.002 (18.320) | 87.286 (25.114)
  Weeks 44-52: number analyzed (Participants) | 331 | 371
  Weeks 44-52 | 89.421 (24.267) | 86.914 (25.366)
  Weeks 96-104: number analyzed (Participants) | 254 | 318
  Weeks 96-104 | 88.858 (24.708) | 83.543 (30.296)

17. Secondary Outcome: Percentage of Hb Values Within 10.0 to 12.0 g/dL in Weeks 28 to 36, 44 to 52, and 96 to 104 Without Use of Rescue Therapy
Description: Percentage for each participant was calculated as Number of Hb values within 10.0-12.0 g/dL / Total number of Hb values*100 in weeks 28 to 36, 44 to 52 and 96 to 104 without use of rescue therapy within 6 weeks prior to and during the 8 week evaluation period.
Time Frame: Weeks 28-36, 44-52 and 96-104
Population: The analysis population was the FAS.
Measure: Mean (Standard Deviation); unit: percentage of Hb values
Arm/Group | Roxadustat | ESA (Erythropoiesis-Stimulating Agent)
Number analyzed (Participants) | 413 | 420
percentage of Hb values
  Weeks 28-36: number analyzed (Participants) | 364 | 393
  Weeks 28-36 | 76.326 (28.175) | 76.098 (28.991)
  Weeks 44-52: number analyzed (Participants) | 331 | 371
  Weeks 44-52 | 75.891 (31.047) | 74.634 (30.589)
  Weeks 96-104: number analyzed (Participants) | 254 | 318
  Weeks 96-104 | 76.522 (30.378) | 73.690 (33.040)

18. Secondary Outcome: Number of Hospitalizations
Description: The number of hospitalizations per participant were calculated during the Efficacy Emergent Period. The Efficacy Emergent Period was defined as the evaluation period from the Analysis date of first dose intake up to EOT Visit or last non-missing Hb assessment (for participants who died during the treatment period). It included all Non-Hemodialysis (HD) hospitalizations. The HD days were not counted as hospitalizations, even when performed overnight.
Time Frame: Baseline to End of Treatment (EOT) (Up to week 104)
Population: The analysis population was the FAS, with participants who had available data.
Measure: Mean (Standard Deviation); unit: Hospitalizations
Arm/Group | Roxadustat | ESA (Erythropoiesis-Stimulating Agent)
Number analyzed (Participants) | 413 | 420
Hospitalizations | 0.9 (1.3) | 0.9 (1.5)

19. Secondary Outcome: Number of Days of Hospitalization Per Year
Description: The number of days of hospitalizations per year was calculated as the sum of the durations of all non-HD hospitalizations in days (Date of discharge - Date of admission + 1)] / (duration of efficacy emergent period in days / 365.25). In case of missing dates, the hospitalization duration was imputed by the average duration per stay derived from the participants with non-missing duration within the same treatment group.
Time Frame: Baseline to EOT (Up to week 104)
Population: The analysis population was the FAS, with participants who had available data.
Measure: Mean (Standard Deviation); unit: Days per year
Arm/Group | Roxadustat | ESA (Erythropoiesis-Stimulating Agent)
Number analyzed (Participants) | 413 | 420
Days per year | 12.186 (34.121) | 7.868 (22.948)

20. Secondary Outcome: Time to First Hospitalization
Description: Time to first hospitalization in years was defined in years as: (First event date during the Efficacy Emergent Period - Analysis date of First dose intake +1)/365.25, and the 'First event date' was defined as 'Date of first Admission and 'Analysis Date of first dose intake. For participants without hospitalization, the time to censoring was calculated as: (Date of End of Efficacy Emergent Period - Analysis Date of first dose intake + 1) / 365.25. Date of End of Efficacy Emergent Period was defined as as the treatment period up to the EOT visit. For participants who have experienced more than one hospitalization, only their first event following study treatment was used. Data reported was analyzed by Kaplan-Meier estimate for cumulative proportion and the 95% confidence interval was calculated with Greenwood's formula.
Time Frame: Baseline to EOT (Up to week 104)
Population: The analysis population was the FAS.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Roxadustat | ESA (Erythropoiesis-Stimulating Agent)
Number analyzed (Participants) | 413 | 420
Percentage of participants
  Year 0.5 | 19.4 [15.5 to 23.3] | 18.3 [14.6 to 22.0]
  Year 1 | 32.0 [27.3 to 36.6] | 32.7 [28.2 to 37.3]
  Year 1.5 | 43.5 [38.5 to 48.6] | 41.9 [37.0 to 46.7]
  Year 2 | 52.6 [47.5 to 57.8] | 48.3 [43.3 to 53.3]
Statistical Analysis 1: Comparison: Roxadustat vs ESA (Erythropoiesis-Stimulating Agent); Hazard Ratio was calculated using stratified Cox Proportional Hazards regression stratifying on region, CV history, previous ESA treatment and adjusting on Hb at baseline as continuous covariate. Superiority was declared if the upper bound of the 95% CI was below 1.0; Test type: Superiority; p = 0.164, Regression, Cox — p-value for superiority test based on 2-sided significance level; Hazard Ratio (HR) = 1.154, 95% CI 2-sided [0.943 to 1.411]

21. Secondary Outcome: Time to First Use of Rescue Therapy
Description: Rescue therapy was defined as red blood cell (RBC) transfusion for both treatment groups and ESA for roxadustat participants. Only rescue medication that was started during the study treatment and up to end of efficacy emergent period was taken into account and considered as use of rescue medication. For participants who have experienced more than one use of rescue therapy, only their first event following study treatment was used. Data reported was analyzed by Kaplan-Meier estimate for cumulative proportion and the 95% confidence interval was calculated with Greenwood's formula.
Time Frame: Baseline to EOT (Up to week 104)
Population: The analysis population was the FAS.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Roxadustat | ESA (Erythropoiesis-Stimulating Agent)
Number analyzed (Participants) | 413 | 420
Percentage of participants
  Year 0.5 | 3.9 [2.0 to 5.8] | 3.2 [1.5 to 4.8]
  Year 1 | 8.2 [5.4 to 11.1] | 8.4 [5.6 to 11.1]
  Year 1.5 | 11.4 [8.1 to 14.8] | 10.9 [7.8 to 14.0]
  Year 2 | 12.8 [9.3 to 16.4] | 14.4 [10.8 to 18.0]
Statistical Analysis 1: Comparison: Roxadustat vs ESA (Erythropoiesis-Stimulating Agent); [analysis description as in outcome 20, analysis 1]; Test type: Superiority; p = 0.917, Regression, Cox; Hazard Ratio (HR) = 0.979, 95% CI 2-sided [0.656 to 1.462]

22. Secondary Outcome: Time to First RBC Transfusion
Description: For participants who have experienced more than one RBC transfusion, only their first event following study treatment was used. For RBC transfusions, when the number of units was not given but the volume transfused was, the number of units were estimated by volume transfused/250 mL (for transfusion of packed cell units) or volume transfused/500 mL (for transfusion of full blood). Data reported was analyzed by Kaplan-Meier estimate for cumulative proportion and the 95% confidence interval was calculated with Greenwood's formula.
Time Frame: Baseline to EOT (Up to week 104)
Population: The analysis population was the FAS.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Roxadustat | ESA (Erythropoiesis-Stimulating Agent)
Number analyzed (Participants) | 413 | 420
Percentage of participants
  Year 0.5 | 3.6 [1.8 to 5.5] | 3.2 [1.5 to 4.8]
  Year 1 | 7.4 [4.7 to 10.1] | 8.4 [5.6 to 11.1]
  Year 1.5 | 10.0 [6.9 to 13.2] | 10.9 [7.8 to 14.0]
  Year 2 | 11.4 [8.0 to 14.9] | 14.4 [10.8 to 18.0]
Statistical Analysis 1: Comparison: Roxadustat vs ESA (Erythropoiesis-Stimulating Agent); Hazard Ratio was calculated using stratified Cox Proportional Hazards regression stratifying on region, CV history, previous ESA treatment, and adjusting on Hb at baseline as continuous covariate. Superiority was declared if the upper bound of the 95% CI was below 1.0; Test type: Superiority; p = 0.501, Regression, Cox — p-value for superiority test based on 2-sided significance level; Hazard Ratio (HR) = 0.867, 95% CI 2-sided [0.573 to 1.313]

23. Secondary Outcome: Mean Monthly Number of RBC Packs Per Participant
Description: During efficacy emergent period, the mean monthly number of RBC packs was calculated as the sum of blood volume and units transfused between the first dose and up to the last dose in the period divided by duration of efficacy emergent period (in days) divided by 28 days. Participants without medication records of RBC have their number of RBC packs and volume set to 0.
Time Frame: Baseline to EOT (Up to week 104)
Population: The analysis population was the FAS.
Measure: Least Squares Mean (95% Confidence Interval); unit: RBC packs per month
Arm/Group | Roxadustat | ESA (Erythropoiesis-Stimulating Agent)
Number analyzed (Participants) | 413 | 420
RBC packs per month | 0.026 [0.01 to 0.04] | 0.032 [0.02 to 0.05]
Statistical Analysis 1: Comparison: Roxadustat vs ESA (Erythropoiesis-Stimulating Agent); The model included treatment arm, region, CV History, previous ESA treatment as categorical variables and baseline Hb as continuous variable; Test type: Superiority; p = 0.507, ANCOVA — p-value for superiority test based on 2-sided significance level; LSM Difference = -0.006, 95% CI 2-sided [-0.02 to 0.01]

24. Secondary Outcome: Mean Monthly Volume of RBC Transfusion Per Participant
Description: During Efficacy Emergent Period, the mean monthly volume of blood transfused was calculated as the sum of blood volume and units transfused between the first dose and up to the last dose in the period divided by duration of efficacy emergent period (in days) divided by 28 days. The Efficacy Emergent Period was defined as the evaluation period from the Analysis date of first dose intake up to EOT Visit or last non-missing Hb assessment (for participants who died during the treatment period).
Time Frame: Baseline to EOT (Up to week 104)
Population: The analysis population was the FAS.
Measure: Least Squares Mean (95% Confidence Interval); unit: mL per month
Arm/Group | Roxadustat | ESA (Erythropoiesis-Stimulating Agent)
Number analyzed (Participants) | 413 | 420
mL per month | 6.061 [2.82 to 9.30] | 5.929 [2.74 to 9.12]
Statistical Analysis 1: Comparison: Roxadustat vs ESA (Erythropoiesis-Stimulating Agent); [analysis description as in outcome 23, analysis 1]; Test type: Superiority; p = 0.949, ANCOVA; LSM Difference = 0.132, 95% CI 2-sided [-3.90 to 4.16]

25. Secondary Outcome: Time to First Use of IV Iron Supplementation
Description: For participants who have received more than one IV iron, only their first event following study treatment was used. Data reported was analyzed by Kaplan-Meier estimate for cumulative proportion and the 95% confidence interval was calculated with Greenwood's formula.
Time Frame: Baseline to EOT (Up to week 104)
Population: The analysis population was the FAS.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Roxadustat | ESA (Erythropoiesis-Stimulating Agent)
Number analyzed (Participants) | 413 | 420
Percentage of participants
  Year 0.5 | 11.2 [8.1 to 14.3] | 33.5 [29.0 to 38.1]
  Year 1 | 17.4 [13.5 to 21.2] | 44.1 [39.3 to 49.0]
  Year 1.5 | 23.6 [19.1 to 28.1] | 55.0 [50.1 to 59.9]
  Year 2 | 33.3 [26.0 to 40.7] | 59.3 [54.4 to 64.3]
Statistical Analysis 1: Comparison: Roxadustat vs ESA (Erythropoiesis-Stimulating Agent); [analysis description as in outcome 20, analysis 1]; Test type: Superiority; p < 0.001, Regression, Cox; Hazard Ratio (HR) = 0.368, 95% CI 2-sided [0.291 to 0.465]

26. Secondary Outcome: Mean Monthly Intravenous (IV) Iron Per Participant During Weeks 37-52 and Weeks 53-104
Description: Participants with no or missing medication records of IV Iron had their monthly IV Iron use set to 0 mg.
Time Frame: Weeks 37-52 and weeks 53-104
Population: The analysis population was the FAS.
Measure: Least Squares Mean (95% Confidence Interval); unit: mg per month
Arm/Group | Roxadustat | ESA (Erythropoiesis-Stimulating Agent)
Number analyzed (Participants) | 413 | 420
mg per month
  Weeks 37-52 | 34.9 [20.9 to 48.9] | 70.0 [56.9 to 83.2]
  Weeks 53-104 | 49.5 [31.0 to 67.9] | 98.1 [81.1 to 115.2]
Statistical Analysis 1: Comparison: Roxadustat vs ESA (Erythropoiesis-Stimulating Agent); Weeks 37-52 - Participants with no or missing medication records of IV Iron had their monthly IV Iron use set to 0 mg. The model includes treatment arm, region, CV History, previous ESA treatment as categorical variables and baseline Hb as continuous variable; Test type: Superiority; p < 0.001, ANCOVA; LSM Difference = -35.1, 95% CI 2-sided [-51.8 to -18.4]
Statistical Analysis 2: Comparison: Roxadustat vs ESA (Erythropoiesis-Stimulating Agent); Weeks 53-104 - Participants with no or missing medication records of IV Iron had their monthly IV Iron use set to 0 mg. The model includes treatment arm, region, CV History, previous ESA treatment as categorical variables and baseline Hb as continuous variable; Test type: Superiority; p < 0.001, ANCOVA; LSM Difference = -48.7, 95% CI 2-sided [-70.3 to -27.0]

27. Secondary Outcome: Percentage of Participants With Oral Iron Use Only
Description: Percentage of participants with/without IV iron only was calculated based on total number of participants within the Efficacy Emergent Period. The Efficacy Emergent Period is defined as the evaluation period from the Analysis date of first dose intake up to EOT Visit or last non-missing Hb assessment (for participants who died during the treatment period).
Time Frame: Baseline to EOT (Up to week 104)
Population: The analysis population was the FAS.
Measure: Number; unit: Percentage of participants
Arm/Group | Roxadustat | ESA (Erythropoiesis-Stimulating Agent)
Number analyzed (Participants) | 413 | 420
Percentage of participants | 31.0 | 11.7

28. Secondary Outcome: Change From BL to Each Post-dosing Study Visit in Total Cholesterol
Description: Baseline assessment was the assessment from Day 1 visit. If baseline value was missing, then the latest screening period value was used as the baseline regardless of fasting status.
Time Frame: Baseline and weeks 8, 28, 52, 104
Population: The analysis population was the FAS.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Roxadustat | ESA (Erythropoiesis-Stimulating Agent)
Number analyzed (Participants) | 413 | 420
mmol/L
  Change from BL to Week 8: number analyzed (Participants) | 392 | 411
  Change from BL to Week 8 | -0.608 (0.889) | -0.105 (0.712)
  Change from BL to Week 28: number analyzed (Participants) | 364 | 393
  Change from BL to Week 28 | -0.641 (0.960) | -0.135 (0.805)
  Change from BL to Week 52: number analyzed (Participants) | 318 | 362
  Change from BL to Week 52 | -0.803 (1.027) | -0.241 (0.906)
  Change from BL to Week 104: number analyzed (Participants) | 247 | 307
  Change from BL to Week 104 | -0.904 (1.053) | -0.277 (1.002)

29. Secondary Outcome: Change From BL to Each Post-dosing Study Visit in LDL-C/High-density Lipoprotein Cholesterol (HDL-C) Ratio
Description: Baseline was defined as the value on Day 1. If baseline value was missing, the latest value prior to first study drug administration was used regardless of fasting.
Time Frame: Baseline and weeks 8, 28, 52, 104
Population: The analysis population was the FAS.
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Roxadustat | ESA (Erythropoiesis-Stimulating Agent)
Number analyzed (Participants) | 413 | 420
Ratio
  Change from BL to Week 8: number analyzed (Participants) | 390 | 411
  Change from BL to Week 8 | -0.245 (0.818) | -0.060 (0.726)
  Change from BL to Week 28: number analyzed (Participants) | 362 | 393
  Change from BL to Week 28 | -0.155 (1.046) | -0.057 (0.922)
  Change from BL to Week 52: number analyzed (Participants) | 317 | 361
  Change from BL to Week 52 | -0.345 (0.904) | -0.078 (0.886)
  Change from BL to Week 104: number analyzed (Participants) | 246 | 307
  Change from BL to Week 104 | -0.261 (1.167) | -0.013 (1.048)

30. Secondary Outcome: Change From BL to Each Postdosing Study Visit in Non-HDL Cholesterol
Description: as for outcome 29
Time Frame: Baseline and weeks 8, 28, 52, 104
Population: The analysis population was the FAS.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Roxadustat | ESA (Erythropoiesis-Stimulating Agent)
Number analyzed (Participants) | 413 | 420
mmol/L
  Change from BL to Week 8: number analyzed (Participants) | 388 | 404
  Change from BL to Week 8 | -0.518 (0.823) | -0.107 (0.701)
  Change from BL to Week 28: number analyzed (Participants) | 360 | 391
  Change from BL to Week 28 | -0.540 (0.907) | -0.127 (0.789)
  Change from BL to Week 52: number analyzed (Participants) | 314 | 360
  Change from BL to Week 52 | -0.700 (0.965) | -0.229 (0.886)
  Change from BL to Week 104: number analyzed (Participants) | 245 | 304
  Change from BL to Week 104 | -0.788 (1.024) | -0.240 (1.010)

31. Secondary Outcome: Change From BL to Each Postdosing Study Visit in Apolipoproteins A1 (ApoA1)
Description: as for outcome 29
Time Frame: Baseline and weeks 8, 28, 52, 104
Population: The analysis population was the FAS.
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Roxadustat | ESA (Erythropoiesis-Stimulating Agent)
Number analyzed (Participants) | 413 | 420
g/L
  Change from BL to Week 8: number analyzed (Participants) | 394 | 415
  Change from BL to Week 8 | -0.114 (0.197) | -0.006 (0.172)
  Change from BL to Week 28: number analyzed (Participants) | 367 | 393
  Change from BL to Week 28 | -0.113 (0.217) | -0.012 (0.193)
  Change from BL to Week 52: number analyzed (Participants) | 320 | 366
  Change from BL to Week 52 | -0.097 (0.230) | -0.013 (0.195)
  Change from BL to Week 104: number analyzed (Participants) | 246 | 309
  Change from BL to Week 104 | -0.097 (0.220) | -0.012 (0.196)

32. Secondary Outcome: Change From BL to Each Postdosing Study Visit in Apolipoproteins B (ApoB)
Description: as for outcome 29
Time Frame: Baseline and weeks 8, 28, 52, 104
Population: The analysis population was the FAS.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Roxadustat | ESA (Erythropoiesis-Stimulating Agent)
Number analyzed (Participants) | 413 | 420
mg/dL
  Change from BL to Week 8: number analyzed (Participants) | 394 | 415
  Change from BL to Week 8 | -11.03 (18.49) | 1.00 (14.34)
  Change from BL to Week 28: number analyzed (Participants) | 366 | 393
  Change from BL to Week 28 | -11.18 (20.39) | -0.12 (16.91)
  Change from BL to Week 52: number analyzed (Participants) | 320 | 366
  Change from BL to Week 52 | -13.18 (20.67) | -0.01 (18.88)
  Change from BL to Week 104: number analyzed (Participants) | 246 | 309
  Change from BL to Week 104 | -13.50 (24.94) | -0.01 (20.00)

33. Secondary Outcome: Change From BL to Each Postdosing Study Visit in ApoB/ApoA1 Ratio
Description: Baseline was defined as the value on Day 1. If baseline value was missing, the latest value prior to first study drug administration was used.
Time Frame: Baseline and weeks 8, 28, 52, 104
Population: The analysis population was the FAS.
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Roxadustat | ESA (Erythropoiesis-Stimulating Agent)
Number analyzed (Participants) | 413 | 420
Ratio
  Change from BL to Week 8: number analyzed (Participants) | 393 | 415
  Change from BL to Week 8 | -0.037 (0.147) | 0.013 (0.141)
  Change from BL to Week 28: number analyzed (Participants) | 365 | 392
  Change from BL to Week 28 | -0.034 (0.177) | 0.002 (0.148)
  Change from BL to Week 52: number analyzed (Participants) | 318 | 365
  Change from BL to Week 52 | -0.051 (0.191) | 0.007 (0.164)
  Change from BL to Week 104: number analyzed (Participants) | 246 | 309
  Change from BL to Week 104 | -0.062 (0.210) | 0.007 (0.201)

34. Secondary Outcome: Number of Participants With Mean LDL Cholesterol < 100 mg/dL Over Weeks 12 to 28
Description: Missing category for Fasting Only includes non-fasting participants and the participants with missing values.
Time Frame: Weeks 12 to 28
Population: The analysis population was the FAS.
Measure: Number; unit: Number of participants
Arm/Group | Roxadustat | ESA (Erythropoiesis-Stimulating Agent)
Number analyzed (Participants) | 413 | 420
Number of participants
  Yes [Regardless of Fasting Status] | 275 | 231
  No [Regardless of Fasting Status] | 119 | 181
  Missing [Regardless of Fasting Status] | 19 | 8
  Yes [Fasting Only] | 111 | 85
  No [Fasting Only] | 61 | 80
  Missing [Fasting Only] | 241 | 255

35. Secondary Outcome: Number of Participants With CKD Who Achieved Antihypertensive Treatment Goal
Description: Achieved antihypertensive treatment goal was defined as SBP < 140 mmHg and DBP < 90 mmHg over an evaluation period based on the average of available values in weeks 12-28 (pre-dialysis).
Time Frame: Weeks 12 to 28
Population: The analysis population was the FAS.
Measure: Number; unit: Number of participants
Arm/Group | Roxadustat | ESA (Erythropoiesis-Stimulating Agent)
Number analyzed (Participants) | 413 | 420
Number of participants
  Antihypertensive Treatment Achievement - Yes | 264 | 261
  Antihypertensive Treatment Achievement - No | 130 | 149
  Antihypertensive Treatment Achievement-Missing | 19 | 10

36. Secondary Outcome: Change From BL to the Average of Weeks 12 to 28 in SF-36 Physical Component Score (PCS)
Description: Baseline SF-36 PCS was defined as the SF-36 PCS value on Day 1. SF-36 contains 36-item that measures 8 scales with scores ranging from 0-100: physical functioning (PF); role limitations due to physical health problems (RP); bodily pain (BP); social functioning (SF); general health perceptions (GH); role limitations due to emotional problems (RE); vitality, energy or fatigue (VT); and mental health (MH). These scores are normed to the US population (norm-based scoring had very little impact on results when data was collected in Western European countries) to have a mean of 50 and standard deviation of 10. The PCS was calculated based on all 8 scales and ranges from 5.02-79.78. For each of these above scales, higher scores always indicating better health status.
Time Frame: Baseline and weeks 12 to 28
Population: The analysis population was the FAS.
Measure: Least Squares Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | Roxadustat | ESA (Erythropoiesis-Stimulating Agent)
Number analyzed (Participants) | 384 | 404
Units on a scale | 0.560 [-0.029 to 1.148] | 0.039 [-0.528 to 0.605]
Statistical Analysis 1: Comparison: Roxadustat vs ESA (Erythropoiesis-Stimulating Agent); The model includes treatment, visit, visit by treatment interaction, Previous ESA Treatment, region and history of CV disease as fixed class factors and baseline SF-36 PCS, baseline Hb, as continuous covariates; Test type: Superiority; p = 0.161, Mixed Models Analysis — p-value for superiority test based on 2-sided significance level; LSM Difference = 0.521, 95% CI 2-sided [-0.208 to 1.250]

37. Secondary Outcome: Change From BL to the Average of Weeks 12 to 28 in Anemia Subscale (AnS) ("Additional Concerns") of Functional Assessment of Cancer Therapy-Anemia (FACT-An) Score
Description: Baseline FACT-An AnS was defined as the FACT-An AnS value on Day 1. Together with the Functional Assessment of Cancer Therapy - General (FACT-G), the Anemia Subscale (AnS) is referred to as the FACT-An Total. The AnS scale contains 13 fatigue specific items (the Fatigue Score) plus 7 items related to anemia. The Anemia AnS score range is 0 to 80. For the above score, a higher score indicates better QoL.
Time Frame: Baseline and weeks 12 to 28
Population: The analysis population was the FAS.
Measure: Least Squares Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | Roxadustat | ESA (Erythropoiesis-Stimulating Agent)
Number analyzed (Participants) | 384 | 403
Units on a scale | 0.400 [-0.624 to 1.424] | 0.274 [-0.709 to 1.257]
Statistical Analysis 1: Comparison: Roxadustat vs ESA (Erythropoiesis-Stimulating Agent); The model includes treatment, visit, visit by treatment interaction, Previous ESA Treatment, region and history of CV disease as fixed class factors and baseline FACT-An Ans, baseline Hb, as continuous covariates; Test type: Superiority; p = 0.845, Mixed Models Analysis — p-value for superiority test based on 2-sided significance level; LSM Difference = 0.126, 95% CI 2-sided [-1.135 to 1.387]

38. Secondary Outcome: Change From BL to the Average Value of Weeks 12 to 28 in Total FACT-An Score
Description: Baseline FACT-An Total Score was defined on Day 1. Total Fact-An score is composed of FACT-G and Ans scales. FACT-G contains 27 items that cover four dimensions of well-being: physical (PWB) - 7 items, functional (FWB) - 7 items, social/family (SWB) - 7 items, and emotional (EWB) - 6 items. The AnS scale contains 13 fatigue specific items (the Fatigue Score) plus 7 items related to anemia. The total score is obtained by summation of the scores from PWB, SWB, EWB, FWB and AnS. The FACT-An Total Score scale range is 0-188. A higher score indicates better QoL.
Time Frame: Baseline and weeks 12 to 28
Population: The analysis population was the FAS.
Measure: Least Squares Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | Roxadustat | ESA (Erythropoiesis-Stimulating Agent)
Number analyzed (Participants) | 383 | 403
Units on a scale | -0.501 [-2.581 to 1.580] | -0.373 [-2.367 to 1.622]
Statistical Analysis 1: Comparison: Roxadustat vs ESA (Erythropoiesis-Stimulating Agent); [analysis description as in outcome 37, analysis 1]; Test type: Superiority; p = 0.922, Mixed Models Analysis — p-value for superiority test based on 2-sided significance level; LSM Difference = -0.128, 95% CI 2-sided [-2.703 to 2.447]

39. Secondary Outcome: Change From BL to the Average of Weeks 12 to 28 in Euroqol Questionnaire-5 Dimensions 5 Levels (EQ-5D 5L) Visual Analogue Scale (VAS) Score
Description: Baseline assessment was defined as the value on Day 1. The EuroQol Questionnaire -5 Dimensions -5 Levels (EQ-5D-5L) is a self-reported questionnaire, used as a measure of respondents' Health Related Quality of Life (HRQoL) and utility values. The EQ-5D consists of the descriptive system and the visual analogue scale (VAS). The EQ-5D descriptive system comprises 5 dimensions of health: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems, extreme problems. The VAS records the respondent's self rated health status on a graduated (0-100) scale, where the endpoints are labeled 'Best imaginable health state' and 'Worst imaginable health state' with higher scores for higher HRQoL.
Time Frame: Baseline and weeks 12 to 28
Population: The analysis population was the FAS.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Roxadustat | ESA (Erythropoiesis-Stimulating Agent)
Number analyzed (Participants) | 385 | 401
Units on a scale | 3.041 (14.910) | 2.735 (14.477)

40. Secondary Outcome: Percentage of Participants With Improvements Measured by Patients' Global Impression of Change (PGIC)
Description: The PGIC is a patient-rated instrument that measures change in participant's overall status on a 7-point scale ranging from 1 (very much improved) to 7 (very much worse), when compared to the start of treatment. The percentage of participants presented includes very much improved, much improved and minimally improved.
Time Frame: Baseline and weeks 8, 12, 28, 36, 52, 76, 104
Population: The analysis population was the FAS.
Measure: Number; unit: Percentage of participants
Arm/Group | Roxadustat | ESA (Erythropoiesis-Stimulating Agent)
Number analyzed (Participants) | 413 | 420
Percentage of participants
  Week 8 | 59.6 | 49.5
  Week 12 | 65.5 | 49.5
  Week 28 | 62.3 | 57.1
  Week 36 | 60.4 | 56.3
  Week 52 | 57.1 | 55.3
  Week 76 | 61.2 | 51.9
  Week 104 | 61.6 | 51.3

41. Secondary Outcome: Change From BL in Serum Hepcidin
Description: Baseline assessment was assessment from Day 1 visit. If baseline value was missing, the value from screening visit was used. In case of missing data, no imputation rules were applied.
Time Frame: Baseline and weeks 4, 12, 20, 36, 52, 104, and End of Study (EOS - up to 108 weeks)
Population: The analysis population was the FAS, with participants who had available data at baseline.
Measure: Mean (Standard Deviation); unit: µg/L
Arm/Group | Roxadustat | ESA (Erythropoiesis-Stimulating Agent)
Number analyzed (Participants) | 413 | 420
µg/L
  Week 4: number analyzed (Participants) | 387 | 400
  Week 4 | -14.265 (42.393) | -4.265 (33.518)
  Week 12: number analyzed (Participants) | 375 | 391
  Week 12 | -12.298 (41.335) | -6.741 (38.507)
  Week 20: number analyzed (Participants) | 361 | 382
  Week 20 | -15.149 (43.152) | -11.818 (41.596)
  Week 36: number analyzed (Participants) | 332 | 366
  Week 36 | -23.405 (43.033) | -14.530 (43.449)
  Week 52: number analyzed (Participants) | 310 | 357
  Week 52 | -32.709 (42.342) | -17.522 (47.307)
  Week 104: number analyzed (Participants) | 242 | 298
  Week 104 | -40.101 (48.611) | -18.735 (51.632)
  EOS: number analyzed (Participants) | 280 | 320
  EOS | -27.192 (52.169) | -17.664 (51.688)

42. Secondary Outcome: Change From BL in Serum Ferritin
Description: as for outcome 41
Time Frame: Baseline and weeks 4, 8, 12, 20, 28, 36, 44, 52, 60, 68, 76, 84, 92, 100, 104, and EOS (up to 108 weeks)
Population: The analysis population was the FAS.
Measure: Mean (Standard Deviation); unit: pmol/L
Arm/Group | Roxadustat | ESA (Erythropoiesis-Stimulating Agent)
Number analyzed (Participants) | 413 | 420
pmol/L
  Week 4: number analyzed (Participants) | 400 | 408
  Week 4 | -214.64 (824.96) | -141.78 (456.15)
  Week 8: number analyzed (Participants) | 394 | 405
  Week 8 | -245.37 (668.51) | -160.75 (607.39)
  Week 12: number analyzed (Participants) | 389 | 404
  Week 12 | -269.76 (761.24) | -179.47 (586.95)
  Week 20: number analyzed (Participants) | 379 | 396
  Week 20 | -337.94 (645.73) | -246.89 (727.64)
  Week 28: number analyzed (Participants) | 363 | 392
  Week 28 | -427.46 (699.95) | -265.21 (816.64)
  Week 36: number analyzed (Participants) | 343 | 379
  Week 36 | -507.34 (726.61) | -269.26 (855.01)
  Week 44: number analyzed (Participants) | 328 | 371
  Week 44 | -545.14 (668.02) | -323.30 (986.38)
  Week 52: number analyzed (Participants) | 318 | 365
  Week 52 | -615.19 (677.97) | -347.58 (1058.87)
  Week 60: number analyzed (Participants) | 304 | 359
  Week 60 | -622.55 (675.22) | -394.40 (837.81)
  Week 68: number analyzed (Participants) | 293 | 349
  Week 68 | -604.47 (773.19) | -456.16 (1039.18)
  Week 76: number analyzed (Participants) | 283 | 339
  Week 76 | -646.76 (838.76) | -447.70 (967.63)
  Week 84: number analyzed (Participants) | 274 | 333
  Week 84 | -629.31 (1060.24) | -454.44 (1193.43)
  Week 92: number analyzed (Participants) | 258 | 326
  Week 92 | -749.58 (828.32) | -371.64 (1157.18)
  Week 100: number analyzed (Participants) | 250 | 313
  Week 100 | -746.86 (796.74) | -364.78 (1802.37)
  Week 104: number analyzed (Participants) | 248 | 308
  Week 104 | -753.82 (791.12) | -348.70 (1292.49)
  EOS: number analyzed (Participants) | 290 | 323
  EOS | -554.53 (910.01) | -166.94 (2035.26)

43. Secondary Outcome: Change From BL in Transferrin Saturation (TSAT)
Description: as for outcome 41
Time Frame: Baseline and weeks 4, 8, 12, 20, 28, 36, 44, 52, 60, 68, 76, 84, 92, 100, 104 and EOS (up to 108 weeks)
Population: The analysis population was the FAS.
Measure: Mean (Standard Deviation); unit: Percentage of saturation
Arm/Group | Roxadustat | ESA (Erythropoiesis-Stimulating Agent)
Number analyzed (Participants) | 412 | 420
Percentage of saturation
  Week 4: number analyzed (Participants) | 392 | 402
  Week 4 | -4.151 (16.147) | -2.331 (13.178)
  Week 8: number analyzed (Participants) | 383 | 399
  Week 8 | -3.681 (17.062) | -3.128 (14.461)
  Week 12: number analyzed (Participants) | 381 | 397
  Week 12 | -2.643 (17.551) | -3.189 (13.912)
  Week 20: number analyzed (Participants) | 363 | 387
  Week 20 | -3.782 (16.634) | -4.398 (14.444)
  Week 28: number analyzed (Participants) | 356 | 385
  Week 28 | -5.463 (17.798) | -3.829 (15.216)
  Week 36: number analyzed (Participants) | 336 | 372
  Week 36 | -5.351 (17.803) | -4.022 (15.471)
  Week 44: number analyzed (Participants) | 320 | 358
  Week 44 | -6.069 (16.349) | -5.254 (15.144)
  Week 52: number analyzed (Participants) | 313 | 353
  Week 52 | -7.278 (17.244) | -5.788 (14.666)
  Week 60: number analyzed (Participants) | 295 | 348
  Week 60 | -6.997 (16.774) | -5.187 (16.097)
  Week 68: number analyzed (Participants) | 287 | 338
  Week 68 | -7.279 (17.809) | -6.237 (15.934)
  Week 76: number analyzed (Participants) | 275 | 332
  Week 76 | -7.156 (17.682) | -6.623 (16.395)
  Week 84: number analyzed (Participants) | 270 | 331
  Week 84 | -7.867 (17.654) | -5.378 (17.771)
  Week 92: number analyzed (Participants) | 251 | 320
  Week 92 | -6.996 (19.850) | -6.259 (16.605)
  Week 100: number analyzed (Participants) | 248 | 308
  Week 100 | -8.379 (17.809) | -6.354 (17.147)
  Week 104: number analyzed (Participants) | 243 | 299
  Week 104 | -7.650 (17.842) | -5.054 (17.195)
  EOS: number analyzed (Participants) | 283 | 321
  EOS | -5.466 (16.626) | -3.763 (17.813)

44. Secondary Outcome: Change From BL in Glycated Hemoglobin (HbA1c) Level to Weeks 12, 28, 36, 44, 52, 60, 84, 104 and EOS (up to Week 108)
Description: Percentage of change from baseline to each study visit were calculated for HbA1c. Baseline assessment was assessment from Day 1 visit. If baseline value was missing, the value from screening visit was used. In case of missing data, no imputation rules were applied.
Time Frame: Baseline and weeks 12, 28, 36, 44, 52, 60, 84, 104 and EOS (up to 108 weeks)
Population: The analysis population was the FAS, with participants who had available data at baseline.
Measure: Mean (Standard Deviation); unit: percentage of Glycated Hemoglobin
Arm/Group | Roxadustat | ESA (Erythropoiesis-Stimulating Agent)
Number analyzed (Participants) | 413 | 419
percentage of Glycated Hemoglobin
  Week 12: number analyzed (Participants) | 385 | 401
  Week 12 | 0.0009 (0.0071) | -0.0005 (0.0057)
  Week 28: number analyzed (Participants) | 360 | 389
  Week 28 | -0.0004 (0.0067) | -0.0006 (0.0064)
  Week 36: number analyzed (Participants) | 342 | 378
  Week 36 | -0.0001 (0.0065) | -0.0004 (0.0067)
  Week 44: number analyzed (Participants) | 327 | 370
  Week 44 | -0.0001 (0.0069) | -0.0006 (0.0067)
  Week 52: number analyzed (Participants) | 317 | 363
  Week 52 | -0.0001 (0.0070) | -0.0007 (0.0068)
  Week 60: number analyzed (Participants) | 303 | 355
  Week 60 | 0.0000 (0.0080) | -0.0004 (0.0070)
  Week 84: number analyzed (Participants) | 269 | 331
  Week 84 | 0.0003 (0.0072) | 0.0001 (0.0078)
  Week 104: number analyzed (Participants) | 242 | 305
  Week 104 | 0.0000 (0.0075) | -0.0003 (0.0082)
  EOS: number analyzed (Participants) | 286 | 319
  EOS | 0.0011 (0.0076) | 0.0001 (0.0080)

45. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs)
Description: Safety was assessed by evaluation of the following variables: (TEAEs; frequency, severity, seriousness, and relationship to study drug), Vital signs (systolic and diastolic blood pressure, pulse, respiratory rate and weight), Clinical laboratory variables (hematology, biochemistry including liver enzymes and total bilirubin, and urinalysis), Physical examination, 12-lead electrocardiogram (ECG) and Vascular Access Thrombosis. All AEs collected during the Safety Emergent Period were counted as TEAE. The TEAE was defined as an adverse event (AE) if it was observed after starting administration of the roxadustat or ESA. Any clinically significant abnormalities were reported as an AEs. All reported deaths after the first study drug administration and up to 28 days after the Analysis Date of Last Dose and considering last dosing frequency.
Time Frame: Baseline up to EOS (Up to week 108)
Population: The analysis population was the Safety Analysis Set (SAF) which consisted of all randomized participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Roxadustat | ESA (Erythropoiesis-Stimulating Agent)
Number analyzed (Participants) | 414 | 420
Participants
  TEAE | 359 | 361
  Drug-Related TEAE | 77 | 35
  Serious TEAE | 210 | 189
  Drug-Related Serious TEAE | 33 | 10
  TEAE Leading to Death | 67 | 55
  Drug-Related TEAE Leading to Death | 5 | 2
  TEAE Leading to Withdrawal of Treatment | 35 | 16
  Drug-Related TEAE Leading to Withdraw of Treatment | 9 | 1
  TEAE NCI CTC Grades 3 or Higher | 181 | 149
  Death During the Safety Emergent Period | 64 | 51
  Death | 78 | 59

ADVERSE EVENTS:
Time Frame: From first dose of study drug up to End of Study (EOS) (Up to week 108)
Description: The Safety Emergent Period was defined as the evaluation period from the Analysis date of first drug intake up to 28 days after the end of treatment taking into account the different dosing frequencies of the study treatments.
Arm/Group | Roxadustat | ESA (Erythropoiesis-Stimulating Agent)
All-Cause Mortality (participants affected / at risk) | 78/414 | 59/420
Serious Adverse Events (participants affected / at risk) | 210/414 | 189/420
Other Adverse Events (participants affected / at risk) | 210/414 | 209/420
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Roxadustat (N=414) | ESA (Erythropoiesis-Stimulating Agent) (N=420)
Anaemia (Blood and lymphatic system disorders) | 5 (5) | 7 (8)
Hypocoagulable state (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Acute coronary syndrome (Cardiac disorders) | 3 (3) | 3 (3)
Acute left ventricular failure (Cardiac disorders) | 2 (2) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 9 (9) | 11 (13)
Angina pectoris (Cardiac disorders) | 5 (5) | 6 (8)
Angina unstable (Cardiac disorders) | 0 (0) | 2 (4)
Aortic valve stenosis (Cardiac disorders) | 2 (2) | 1 (1)
Arrhythmia (Cardiac disorders) | 0 (0) | 1 (1)
Arteriosclerosis coronary artery (Cardiac disorders) | 1 (1) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 12 (14) | 8 (8)
Atrial flutter (Cardiac disorders) | 1 (1) | 1 (1)
Atrial tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Atrioventricular block (Cardiac disorders) | 0 (0) | 2 (2)
Atrioventricular block complete (Cardiac disorders) | 1 (1) | 0 (0)
Atrioventricular block second degree (Cardiac disorders) | 0 (0) | 1 (1)
Bradycardia (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac arrest (Cardiac disorders) | 4 (4) | 8 (9)
Cardiac failure (Cardiac disorders) | 8 (8) | 9 (9)
Cardiac failure acute (Cardiac disorders) | 3 (3) | 1 (1)
Cardiac failure chronic (Cardiac disorders) | 1 (1) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 5 (5) | 1 (1)
Cardiac fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Cardio-respiratory arrest (Cardiac disorders) | 1 (1) | 2 (3)
Cardiogenic shock (Cardiac disorders) | 2 (2) | 1 (1)
Cardiopulmonary failure (Cardiac disorders) | 3 (3) | 1 (1)
Cardiovascular insufficiency (Cardiac disorders) | 2 (2) | 0 (0)
Coronary artery disease (Cardiac disorders) | 2 (2) | 3 (3)
Coronary artery occlusion (Cardiac disorders) | 1 (1) | 0 (0)
Coronary artery stenosis (Cardiac disorders) | 1 (1) | 2 (2)
Diastolic dysfunction (Cardiac disorders) | 0 (0) | 1 (1)
Hypertensive heart disease (Cardiac disorders) | 0 (0) | 1 (1)
Left ventricular failure (Cardiac disorders) | 1 (1) | 0 (0)
Mitral valve incompetence (Cardiac disorders) | 0 (0) | 1 (1)
Mitral valve stenosis (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 6 (6)
Myocardial ischaemia (Cardiac disorders) | 4 (5) | 4 (4)
Pericarditis (Cardiac disorders) | 1 (1) | 0 (0)
Sinus node dysfunction (Cardiac disorders) | 0 (0) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 5 (5)
Tachyarrhythmia (Cardiac disorders) | 0 (0) | 1 (1)
Tricuspid valve incompetence (Cardiac disorders) | 0 (0) | 1 (1)
Ventricular arrhythmia (Cardiac disorders) | 0 (0) | 1 (2)
Ventricular fibrillation (Cardiac disorders) | 1 (1) | 2 (2)
Hypoacusis (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Hyperparathyroidism secondary (Endocrine disorders) | 3 (3) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 1 (1) | 0 (0)
Toxic goitre (Endocrine disorders) | 1 (1) | 0 (0)
Angle closure glaucoma (Eye disorders) | 0 (0) | 1 (1)
Cataract (Eye disorders) | 0 (0) | 1 (1)
Eye haemorrhage (Eye disorders) | 1 (1) | 1 (1)
Abdominal adhesions (Gastrointestinal disorders) | 0 (0) | 1 (2)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal wall haematoma (Gastrointestinal disorders) | 0 (0) | 1 (1)
Acute abdomen (Gastrointestinal disorders) | 0 (0) | 1 (1)
Anal fissure (Gastrointestinal disorders) | 1 (1) | 0 (0)
Anal fistula (Gastrointestinal disorders) | 1 (1) | 0 (0)
Anal incontinence (Gastrointestinal disorders) | 0 (0) | 1 (1)
Chronic gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Colitis ischaemic (Gastrointestinal disorders) | 0 (0) | 1 (2)
Constipation (Gastrointestinal disorders) | 1 (1) | 2 (3)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 3 (4)
Diverticulum (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diverticulum intestinal (Gastrointestinal disorders) | 0 (0) | 2 (2)
Duodenal ulcer (Gastrointestinal disorders) | 4 (4) | 0 (0)
Erosive duodenitis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Faecaloma (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastritis erosive (Gastrointestinal disorders) | 2 (2) | 2 (2)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 6 (6)
Gastrointestinal ischaemia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal necrosis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ileus paralytic (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal ischaemia (Gastrointestinal disorders) | 1 (1) | 2 (2)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intestinal ulcer perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intra-abdominal haematoma (Gastrointestinal disorders) | 0 (0) | 1 (1)
Large intestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Large intestine perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Mechanical ileus (Gastrointestinal disorders) | 0 (0) | 1 (1)
Melaena (Gastrointestinal disorders) | 1 (1) | 2 (2)
Nausea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Oesophageal ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 3 (3)
Ulcerative gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 (3) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1)
Asthenia (General disorders) | 3 (3) | 1 (1)
Catheter site haematoma (General disorders) | 0 (0) | 1 (1)
Catheter site inflammation (General disorders) | 1 (1) | 0 (0)
Chest pain (General disorders) | 1 (1) | 0 (0)
Chills (General disorders) | 1 (1) | 0 (0)
Complication associated with device (General disorders) | 1 (1) | 1 (1)
Death (General disorders) | 6 (6) | 3 (3)
Device related thrombosis (General disorders) | 3 (5) | 1 (1)
Hyperthermia (General disorders) | 0 (0) | 1 (1)
Impaired healing (General disorders) | 0 (0) | 1 (1)
Malaise (General disorders) | 1 (1) | 1 (1)
Medical device site phlebitis (General disorders) | 1 (2) | 0 (0)
Multiple organ dysfunction syndrome (General disorders) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 1 (1)
Pain (General disorders) | 0 (0) | 2 (2)
Peripheral swelling (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 4 (4) | 4 (5)
Sudden cardiac death (General disorders) | 1 (1) | 1 (1)
Sudden death (General disorders) | 7 (7) | 3 (3)
Vascular stent stenosis (General disorders) | 0 (0) | 1 (1)
Bile duct obstruction (Hepatobiliary disorders) | 1 (1) | 0 (0)
Bile duct stone (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholangitis (Hepatobiliary disorders) | 1 (1) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 3 (3)
Hepatotoxicity (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 (1) | 0 (0)
Jaundice (Hepatobiliary disorders) | 1 (1) | 0 (0)
Anti-neutrophil cytoplasmic antibody positive vasculitis (Immune system disorders) | 0 (0) | 1 (1)
Renal transplant failure (Immune system disorders) | 1 (1) | 0 (0)
Abdominal abscess (Infections and infestations) | 0 (0) | 1 (1)
Abdominal infection (Infections and infestations) | 1 (1) | 0 (0)
Abscess neck (Infections and infestations) | 0 (0) | 1 (1)
Acute hepatitis B (Infections and infestations) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 2 (2) | 1 (1)
Arteriovenous fistula site infection (Infections and infestations) | 3 (3) | 0 (0)
Arthritis bacterial (Infections and infestations) | 2 (2) | 0 (0)
Bacterial sepsis (Infections and infestations) | 0 (0) | 1 (1)
Biliary sepsis (Infections and infestations) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 5 (5) | 3 (3)
Cellulitis (Infections and infestations) | 2 (2) | 1 (1)
Cholecystitis infective (Infections and infestations) | 0 (0) | 1 (1)
Clostridium difficile infection (Infections and infestations) | 1 (1) | 0 (0)
Device related infection (Infections and infestations) | 2 (2) | 3 (4)
Device related sepsis (Infections and infestations) | 3 (3) | 3 (3)
Diabetic gangrene (Infections and infestations) | 2 (2) | 0 (0)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0)
Encephalomyelitis (Infections and infestations) | 1 (1) | 0 (0)
Endocarditis (Infections and infestations) | 2 (3) | 0 (0)
Enterobacter bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Enterococcal sepsis (Infections and infestations) | 0 (0) | 1 (1)
Erysipelas (Infections and infestations) | 1 (1) | 3 (3)
Escherichia bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Escherichia urinary tract infection (Infections and infestations) | 1 (2) | 1 (1)
Fungal oesophagitis (Infections and infestations) | 1 (1) | 0 (0)
Gangrene (Infections and infestations) | 5 (6) | 4 (7)
Gastric ulcer helicobacter (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 6 (6)
Gastrointestinal candidiasis (Infections and infestations) | 1 (1) | 0 (0)
Haematoma infection (Infections and infestations) | 0 (0) | 2 (2)
Incision site infection (Infections and infestations) | 1 (1) | 0 (0)
Infected skin ulcer (Infections and infestations) | 1 (1) | 0 (0)
Infectious colitis (Infections and infestations) | 0 (0) | 2 (2)
Influenza (Infections and infestations) | 2 (2) | 1 (1)
Intervertebral discitis (Infections and infestations) | 1 (1) | 0 (0)
Liver abscess (Infections and infestations) | 1 (1) | 0 (0)
Localised infection (Infections and infestations) | 0 (0) | 2 (2)
Lower respiratory tract infection (Infections and infestations) | 2 (2) | 0 (0)
Lung abscess (Infections and infestations) | 1 (1) | 0 (0)
Medical device site joint infection (Infections and infestations) | 1 (1) | 0 (0)
Osteomyelitis (Infections and infestations) | 1 (2) | 0 (0)
Osteomyelitis bacterial (Infections and infestations) | 0 (0) | 1 (1)
Pancreatitis bacterial (Infections and infestations) | 1 (1) | 0 (0)
Penile abscess (Infections and infestations) | 0 (0) | 1 (1)
Periodontitis (Infections and infestations) | 0 (0) | 1 (1)
Peritonitis (Infections and infestations) | 10 (15) | 3 (4)
Peritonitis bacterial (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 15 (15) | 21 (22)
Pneumonia pneumococcal (Infections and infestations) | 1 (1) | 0 (0)
Postoperative wound infection (Infections and infestations) | 1 (1) | 0 (0)
Pseudomonal sepsis (Infections and infestations) | 1 (1) | 0 (0)
Pyelonephritis (Infections and infestations) | 1 (1) | 0 (0)
Pyelonephritis acute (Infections and infestations) | 1 (1) | 1 (1)
Pyelonephritis chronic (Infections and infestations) | 2 (2) | 0 (0)
Pyonephrosis (Infections and infestations) | 1 (1) | 0 (0)
Renal abscess (Infections and infestations) | 1 (1) | 0 (0)
Renal cyst infection (Infections and infestations) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 2 (2)
Respiratory tract infection bacterial (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 8 (8) | 9 (9)
Sepsis syndrome (Infections and infestations) | 1 (1) | 0 (0)
Septic shock (Infections and infestations) | 1 (1) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Skin infection (Infections and infestations) | 1 (1) | 0 (0)
Soft tissue infection (Infections and infestations) | 0 (0) | 1 (1)
Staphylococcal bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Staphylococcal sepsis (Infections and infestations) | 3 (3) | 2 (2)
Streptococcal sepsis (Infections and infestations) | 0 (0) | 1 (1)
Subcutaneous abscess (Infections and infestations) | 1 (1) | 0 (0)
Systemic infection (Infections and infestations) | 1 (1) | 0 (0)
Tracheobronchitis (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1)
Urinary tract infection (Infections and infestations) | 4 (4) | 0 (0)
Urinary tract infection bacterial (Infections and infestations) | 1 (1) | 2 (2)
Urinary tract infection enterococcal (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection pseudomonal (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection staphylococcal (Infections and infestations) | 1 (1) | 0 (0)
Urosepsis (Infections and infestations) | 1 (1) | 2 (2)
Viral upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Arteriovenous fistula aneurysm (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Arteriovenous fistula occlusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Arteriovenous fistula site complication (Injury, poisoning and procedural complications) | 6 (7) | 5 (5)
Arteriovenous fistula site haemorrhage (Injury, poisoning and procedural complications) | 2 (3) | 1 (1)
Arteriovenous fistula thrombosis (Injury, poisoning and procedural complications) | 29 (37) | 15 (18)
Arteriovenous graft site haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Arteriovenous graft site stenosis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Arteriovenous graft thrombosis (Injury, poisoning and procedural complications) | 1 (1) | 2 (5)
Back injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Comminuted fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Facial bones fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (2)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 6 (6)
Femoral neck fracture (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 2 (2) | 5 (5)
Graft thrombosis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Ligament rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Lip injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Lower limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Poisoning (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post procedural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Post procedural inflammation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Procedural complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Pubis fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Shunt aneurysm (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Shunt malfunction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Shunt occlusion (Injury, poisoning and procedural complications) | 2 (5) | 1 (1)
Shunt stenosis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Shunt thrombosis (Injury, poisoning and procedural complications) | 1 (1) | 4 (5)
Skin injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Skin wound (Injury, poisoning and procedural complications) | 1 (2) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Spinal fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Subdural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Tibia fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Ulna fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Upper limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Vascular access malfunction (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Vascular access site haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (2)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Wound (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Blood potassium increased (Investigations) | 1 (1) | 0 (0)
Electrocardiogram abnormal (Investigations) | 0 (0) | 1 (1)
Cachexia (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Diabetes mellitus (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Fluid overload (Metabolism and nutrition disorders) | 1 (1) | 2 (3)
Fluid retention (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 2 (3) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 4 (4) | 3 (3)
Hypervolaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Metabolic acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Fistula discharge (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Joint contracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Mobility decreased (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Sarcopenia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (3) | 2 (2)
Benign lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Benign renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Carcinoid tumour pulmonary (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Colorectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Colorectal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Endometrial adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Haemangioma of bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Hypopharyngeal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Kidney angiomyolipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 2 (2)
Malignant neoplasm of choroid (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Ovarian neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Parathyroid tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Penile cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Refractory anaemia with an excess of blasts (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Carotid artery stenosis (Nervous system disorders) | 0 (0) | 1 (2)
Carpal tunnel syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Cerebellar infarction (Nervous system disorders) | 0 (0) | 1 (1)
Cerebral arteriosclerosis (Nervous system disorders) | 0 (0) | 1 (1)
Cerebral artery occlusion (Nervous system disorders) | 0 (0) | 1 (1)
Cerebral haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral infarction (Nervous system disorders) | 0 (0) | 4 (5)
Cerebral ischaemia (Nervous system disorders) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 3 (3) | 1 (1)
Cerebrovascular disorder (Nervous system disorders) | 0 (0) | 1 (1)
Cognitive disorder (Nervous system disorders) | 1 (1) | 0 (0)
Coma (Nervous system disorders) | 1 (1) | 2 (2)
Disturbance in attention (Nervous system disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Embolic cerebral infarction (Nervous system disorders) | 0 (0) | 1 (1)
Encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Epilepsy (Nervous system disorders) | 0 (0) | 1 (1)
Epileptic encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Generalised tonic-clonic seizure (Nervous system disorders) | 1 (2) | 0 (0)
Haemorrhage intracranial (Nervous system disorders) | 1 (1) | 0 (0)
Haemorrhagic stroke (Nervous system disorders) | 0 (0) | 1 (1)
Hypoxic-ischaemic encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Idiopathic partial epilepsy (Nervous system disorders) | 1 (1) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 1 (1) | 1 (1)
Lethargy (Nervous system disorders) | 0 (0) | 1 (1)
Loss of consciousness (Nervous system disorders) | 2 (2) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 2 (2)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 2 (2)
Vascular dementia (Nervous system disorders) | 0 (0) | 1 (1)
Vertigo CNS origin (Nervous system disorders) | 1 (1) | 0 (0)
Device dislocation (Product Issues) | 0 (0) | 1 (1)
Device failure (Product Issues) | 2 (2) | 0 (0)
Device malfunction (Product Issues) | 4 (5) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 2 (2)
Delirium (Psychiatric disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Disorientation (Psychiatric disorders) | 0 (0) | 1 (1)
Fear of falling (Psychiatric disorders) | 1 (1) | 0 (0)
Mental disorder due to a general medical condition (Psychiatric disorders) | 1 (1) | 0 (0)
Organic brain syndrome (Psychiatric disorders) | 0 (0) | 1 (1)
Calculus urinary (Renal and urinary disorders) | 1 (1) | 0 (0)
Chronic kidney disease (Renal and urinary disorders) | 1 (1) | 0 (0)
End stage renal disease (Renal and urinary disorders) | 0 (0) | 2 (2)
Haematuria (Renal and urinary disorders) | 1 (1) | 2 (2)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 2 (3)
Renal cyst ruptured (Renal and urinary disorders) | 1 (1) | 2 (2)
Tubulointerstitial nephritis (Renal and urinary disorders) | 0 (0) | 1 (1)
Urethral perforation (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinoma (Renal and urinary disorders) | 1 (1) | 0 (0)
Ovarian disorder (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Uterine polyp (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Chronic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 4 (4)
Eosinophilic pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 6 (7) | 2 (3)
Pleural thickening (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pulmonary alveolar haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 1 (1)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Pulmonary infarction (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 2 (2)
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Cutaneous vasculitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Diabetic foot (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Ingrowing nail (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Neurodermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash vesicular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin necrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Toxic epidermal necrolysis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Catheter placement (Surgical and medical procedures) | 1 (1) | 0 (0)
Therapy cessation (Surgical and medical procedures) | 1 (1) | 0 (0)
Aortic dissection (Vascular disorders) | 1 (1) | 0 (0)
Aortic stenosis (Vascular disorders) | 0 (0) | 1 (1)
Arterial disorder (Vascular disorders) | 0 (0) | 1 (1)
Circulatory collapse (Vascular disorders) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 4 (5) | 0 (0)
Diabetic vascular disorder (Vascular disorders) | 1 (1) | 0 (0)
Dry gangrene (Vascular disorders) | 1 (1) | 2 (3)
Haematoma (Vascular disorders) | 0 (0) | 3 (3)
Haemorrhage (Vascular disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 10 (10) | 5 (5)
Hypertensive crisis (Vascular disorders) | 3 (4) | 3 (8)
Hypotension (Vascular disorders) | 4 (5) | 1 (3)
Intermittent claudication (Vascular disorders) | 0 (0) | 1 (1)
Lymphoedema (Vascular disorders) | 1 (1) | 0 (0)
Malignant hypertension (Vascular disorders) | 1 (1) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 1 (1) | 1 (1)
Peripheral arterial occlusive disease (Vascular disorders) | 2 (2) | 4 (4)
Peripheral artery occlusion (Vascular disorders) | 0 (0) | 3 (3)
Peripheral artery stenosis (Vascular disorders) | 0 (0) | 1 (1)
Peripheral artery thrombosis (Vascular disorders) | 2 (2) | 0 (0)
Peripheral ischaemia (Vascular disorders) | 2 (2) | 4 (6)
Peripheral vascular disorder (Vascular disorders) | 0 (0) | 1 (1)
Steal syndrome (Vascular disorders) | 1 (1) | 0 (0)
Subclavian artery thrombosis (Vascular disorders) | 1 (1) | 1 (1)
Subclavian vein thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Thrombosis (Vascular disorders) | 1 (2) | 1 (1)
Vasculitis necrotising (Vascular disorders) | 0 (0) | 1 (2)
Venous stenosis (Vascular disorders) | 1 (1) | 1 (5)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Roxadustat (N=414) | ESA (Erythropoiesis-Stimulating Agent) (N=420)
Hyperparathyroidism secondary (Endocrine disorders) | 21 (21) | 16 (17)
Diarrhoea (Gastrointestinal disorders) | 33 (51) | 32 (60)
Nausea (Gastrointestinal disorders) | 27 (29) | 8 (10)
Bronchitis (Infections and infestations) | 29 (38) | 27 (34)
Upper respiratory tract infection (Infections and infestations) | 14 (19) | 21 (29)
Viral upper respiratory tract infection (Infections and infestations) | 28 (61) | 39 (68)
Arteriovenous fistula thrombosis (Injury, poisoning and procedural complications) | 27 (34) | 18 (21)
Iron deficiency (Metabolism and nutrition disorders) | 30 (39) | 51 (64)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 15 (21) | 33 (48)
Headache (Nervous system disorders) | 36 (41) | 29 (39)
Hypertension (Vascular disorders) | 66 (101) | 75 (116)
Hypotension (Vascular disorders) | 30 (40) | 26 (40)

LIMITATIONS AND CAVEATS:
Overall 838 were randomized to receive treatment. Two participants randomized to the pooled ESA treatment group were excluded due to GCP violations and their data was excluded. Total of 836 were considered randomized.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institute and/or Principal Investigator may publish trial data generated at their specific study site after Sponsor publication of the multi-center data. Sponsor must receive a site's manuscript prior to publication for review and comment as specified in the Investigator Agreement.

DOCUMENTS (2):
  • Study Protocol (2017-05-30): https://cdn.clinicaltrials.gov/large-docs/41/NCT02278341/Prot_000.pdf
  • Statistical Analysis Plan (2018-09-10): https://cdn.clinicaltrials.gov/large-docs/41/NCT02278341/SAP_001.pdf